209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | Immunogenicity and safety study of GSK's investigational vaccine (GSK3277511A) when administered in healthy smokers and ex-smokers following receipt of <i>Shingrix</i> vaccine. |
| eTrack study number and<br>Abbreviated Title | 209538 (NTHI MCAT-009) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Amendment 2 Final: 20 May 2020 |

APP 9000058193 Statistical Analysis Plan Template V4 (Effective date: 3June2019)

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | ST OF A | BBREVIA | TIONS | | 6 |
| 1. | DOCU | JMENT H | ISTORY | | 8 |
| 2. | STUD | Y DESIG | N | | 9 |
| 3. | OBJE | CTIVES A | AND ENDPO | INTS | 11 |
| 4. | ANAL | YSIS SET | | | 14 |
| • | 4.1. | | | | |
| | | 4.1.1. | | considerations | |
| | 4.2. | Criteria | | g data from Analysis Sets | |
| | | 4.2.1. | Elimination | from Exposed Set (ES) | 14 |
| | | 4.2.2. | | from Full analysis set (FAS) | |
| | | | 4.2.2.1. | Excluded subjects | 15 |
| | | 4.2.3. | | from Modified full analysis set (mFAS) | |
| | | | 4.2.3.1. | Excluded subjects | 15 |
| | | 4.2.4. | Elimination | from Per-protocol analysis set (PPS) | 16 |
| | | | | Excluded subjects | |
| | | 4.2.5. | | from unsolicited and solicited safety set | |
| | | | | Excluded subjects | |
| | | | | 4.2.5.1.1. Unsolicited safety set | 16 |
| | | | | 4.2.5.1.2. Solicited safety set | 17 |
| 5. | | STATISTICAL ANALYSES | | | |
| | 5.1. Demography | | | | |
| | | 5.1.1. | Analysis of | demographics/baseline characteristics planned | 17 |
| | | 5.1.2. | Additional | considerations | 18 |
| | 5.2. | • | | | |
| | 0.2. | 5.2.1. | | exposure planned in the protocol | |
| | | 5.2.2. | Additional | considerations | 18 |
| | 5.3. | - | | | |
| | | 5.3.1. | | immunogenicity planned in the protocol | |
| | | 5.3.2. | | considerations | |
| | | | | Analysis of humoral response | |
| | | | | Analysis of CMI response | |
| | 5.4. | Analysis | | d reactogenicity | |
| | | 5.4.1. | | safety and reactogenicity planned in the | |
| | | | | | 23 |
| | | 5.4.2. | | considerations | |
| | | | 5.4.2.1. | Analysis of solicited AEs | 23 |
| | | | | Analysis of unsolicited AEs | |
| | | | 5.4.2.3. | Combined analysis of solicited and unsolicited AEs | |
| | | | | Analysis of SAEs and pIMDs | |
| | | | | Other safety analyses | |
| 6 | ANAI | YSIS INT | ERPRETATI | ON | 26 |

| 209538 (NTHI MCAT-009) |
|---------------------------------------|
| Statistical Analysis Plan Amendment 2 |

| | | | | Statistical Analysis Plan Amend | ment 2 |
|---|---|---|---|---|---|
| 7. | | | | <b>)</b> | |
| | 7.1. | | | es | |
| | 7.2. | Statistic | al considera | tions for interim analyses | 27 |
| 8. | CHAN | GES FRO | OM PLANNE | ED ANALYSES | 28 |
| 9. | | | | ERIVATION RULES AND STATISTICAL | |
| | 9.1. | | | | |
| | | 9.1.1. | | -offs for serology results | |
| | 9.2. | 9.1.2.<br>Statistic | | subjects to time-lag groups | |
| | 0.2. | Otationo | ai wearoa | | 20 |
| 10. | | | | | |
| | 10.1. | | | tandard data derivations and statistical methods | |
| | | 10.1.1. | | events to vaccine doses | |
| | | 10.1.2. | | of missing data | |
| | | | | Dates | |
| | | | | Laboratory data | |
| | | | 10.1.2.3. | Daily recording of solicited symptoms | |
| | | | 40.4.0.4 | 10.1.2.3.1. Studies with paper diaries | |
| | | 40.4.0 | 10.1.2.4. | Unsolicited adverse events | |
| | | 10.1.3. | | ration | |
| | | | 10.1.3.1. | Age at vaccination in years | |
| | | | 10.1.3.2. | Body mass index (BMI) | |
| | | | 10.1.3.3. | Numerical serology results | |
| | | | 10.1.3.4. | Geometric mean concentrations (GMCs) | |
| | | | 10.1.3.5.<br>10.1.3.6. | Onset day Duration of events | |
| | | | 10.1.3.0. | Counting rules for combining solicited and | 32 |
| | | | 10.1.3.7. | unsolicited adverse events | 33 |
| | | | 10.1.3.8. | Counting rules for occurrences of solicited | 33 |
| | | | 10.1.5.0. | adverse events | 33 |
| | | 10.1.4. | Display of | decimals | |
| | | 10.1.4. | | Percentages | |
| | | | 10.1.4.1. | Differences in percentages | |
| | | | 10.1.4.3. | Demographic/baseline characteristics statistics | |
| | | | 10.1.4.4. | Serological summary statistics | |
| | | 10.1.5. | | methodology | |
| | | 10.1.0. | | Exact confidence intervals around proportions | |
| | | | 10.1.5.2. | | |
| | | | | around differences in proportions | 35 |
| | | | 10.1.5.3. | Adjusted GMC ratios | |
| | 10.2. | TFL To | <b>)</b> | | 35 |
| | 10.3. | | | hod and minimization algorithm | 35 |
| 11 | REEE | RENCES | | | 37 |
| 10.0 | | | | | |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

# **LIST OF TABLES**

| | | PAGE |
|---------|----------------------------------------------------------|------|
| Table 1 | Study groups, treatment and epochs foreseen in the study | 10 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| igure 1 | Study design overview | 9 |
| Figure 2 | Sequence for evaluating the primary objective in order to control the overall type I error below 2.5% (one-sided) in case all groups reached the number of subjects planned in the PPS | 26 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## LIST OF ABBREVIATIONS

AE Adverse event

ANCOVA Analysis of Covariance

ANOVA Analysis of Variance

CI Confidence Interval

CMI Cell-Mediated Immune

COVID-19 Coronavirus Disease 2019

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

eCRF Electronic Case Report Form

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set

eTMF Electronic Trial Master File

EU/mL ELISA unit per milliliter

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMR Geometric mean ratio

GSK GlaxoSmithKline

LL Lower Limit

LLOQ Lower Limit of Quantification

MedDRA Medical Dictionary for Regulatory Activities

mFAS Modified Full Analysis Set

NA Not Applicable

NI Non-Inferiority

PD Protocol Deviation

## 209538 | Statistical Analysis Plan Amendment 2 20 May 2020 | TMF-1783938 | 2.0

## CONFIDENTIAL

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

PPS Per-Protocol Set

RCD Reverse cumulative distribution

SAE Serious adverse event

SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SDTM Study Data Tabulation Model

SR Study Report

TFL Tables Figures and Listings

ToC Table of Content

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 01 APR 2019 | First version | Protocol Administrative<br>Change 1: 14 DEC<br>2018 |
| 30 JAN 2020 | Amendment 1: • Section 5.3.2.1: update to the permutation test algorithm (recommendation from Center for Biologics Evaluation and Research) | Protocol Administrative<br>Change 1: 14 DEC<br>2018 |
| 20 MAY 2020 | <ul> <li>Amendment 2:</li> <li>Section 3: Objectives and endpoints</li> <li>Section 4.2.4.1: Elimination codes from Per Protocol Set</li> <li>Section 5.3.1: Analysis of immunogenicity planned per protocol</li> <li>Section 5.3.2.1: Analysis of humoral response</li> <li>Section 6: Analysis interpretation</li> </ul> | Protocol Amendment 1:<br>18 MAY 2020 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 2. STUDY DESIGN

Figure 1 Study design overview



BS C = blood sample for cell-mediated immune response; BS H = blood sample for humoral immune responses/assay development from all subjects; C= Call; D = Day; mth(s) = month(s); NA = not applicable; NM = NTHi-Mcat vaccination; RAND = randomization; S = Safety; Sh = *Shingrix* vaccination; V = Visit Notes:

- <sup>1</sup> Groups: Sh NTHi-Mcat 1 (NTHi-Mcat vaccine administered 1 month after *Shingrix* vaccine)
- <sup>2</sup> Groups: Sh\_NTHi-Mcat\_3 (NTHi-Mcat vaccine administered 3 months after *Shingrix* vaccine)
- <sup>3</sup> Groups: Sh NTHi-Mcat 6 (NTHi-Mcat vaccine administered 6 months after *Shingrix* vaccine)
- <sup>4</sup> Patients randomized to the NTHi-Mcat control group will receive the first NTHi-Mcat vaccination at Visit 1 (Day 1) and the second NTHi-Mcat vaccination at Visit 3 (Day 61)
- <sup>5</sup> Blood sample for cell-mediated immune response will be taken from approximately 60 subjects ( ~15 subjects in each group. Refer to Section 5.3.1 of the study protocol for details of the CMI sub-cohort
- <sup>6.</sup> Solicited local and general adverse events reported during a 7-day follow-up period after Dose 1 and after Dose 2 of NTHi-Mcat vaccine, and unsolicited adverse events reported during a 30-day follow-up period after Dose 1 and after Dose 2 of NTHi-Mcat vaccine will be collected
- 7. Safety follow-up

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

- **Primary completion date (PCD):** PCD will be 1 month post-Dose 2 of the NTHi-Mcat investigational vaccine (Day 331, based on Sh\_NTHi-Mcat\_6 treatment group).
- End of Study (EoS): Last subject last visit (Day 661).
- **Study groups:** Approximately 540 eligible subjects who will be randomly assigned to 4 study groups in a (1: 1: 1) ratio (Table 1). Please refer to Section 10.1 of the protocol for details related to the determination of sample size.

Table 1 Study groups, treatment and epochs foreseen in the study

| Study Groups | Number<br>of | Age | Age Treatment name | | ochs<br>ding) |
|---|---|---|---|---|---|
| Study Groups | subjects | (Min-Max) | rreatment name | Epoch 001<br>(open-label) | Epoch 002<br>(open-label) |
| Sh_NTHi-Mcat_1 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| Sh_NTHi-Mcat_3 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| Sh_NTHi-Mcat_6 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| NTHi-Mcat | 135 | 50 – 80 years | NTHi-Mcat | • | • |

- **Treatment allocation:** Subjects will be allocated to a study group using an automated, electronic System Built for Internet Randomization (SBIR). The randomization algorithm will use a minimization procedure accounting for age category (50–59, 60–69, 70–80 years of age), smoking status (current or former smoker), and centre. Minimization factors will have equal weight in the minimization algorithm.
- **Blinding:** open-label.
- **Data collection:** Electronic Case Report Form (eCRF). Telephone contact. Solicited and unsolicited symptoms will be collected using a subject Diary (paper diary [pDiary]).
- Safety monitoring: Subjects will be observed for at least 60 minutes after each NTHi-Mcat vaccination for any immediate reactions. Solicited local and general AEs occurring during a 7-day follow-up period after each NTHi-Mcat vaccination (i.e. the day of vaccination and the 6 subsequent days) and unsolicited AEs occurring during a 30-day follow-up period after each NTHi-Mcat vaccination (i.e. the day of vaccination and the 29 subsequent days), will be reported via diary cards. In addition, subjects will be asked at Phone contacts if there were any safety concerns in the 7-day follow-up period after each NTHi-Mcat vaccination; this information will be recorded via the appropriate section of the eCRF. Finally, safety assessments will be performed during each clinic visit and safety follow-up calls to collect information on AEs leading to withdrawal, serious adverse events (SAEs), SAEs related to study participation or to a concurrent GSK medication/vaccine, pregnancies, potential immune-mediated diseases (pIMDs), throughout the whole study period.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

#### 3. **OBJECTIVES AND ENDPOINTS**

| Objectives | Endpoints |
|---|---|
| P | rimary |
| Confirmatory To demonstrate the non-inferiority (NI) of the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine versus the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine alone. Criterion: | <ul> <li>Humoral immune response</li> <li>Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations 1 month after Dose 2 of NTHi-Mcat vaccine in the Sh_NTHi-Mcat groups (Day 181; Day 241; Day 331) compared to antibody concentrations 1 month after Dose 2 in the NTHi-Mcat group (Day 91).1</li> </ul> |
| <ul> <li>Lower limit (LL) of the 2-sided 95% confidence<br/>interval (CI) of the geometric mean concentration<br/>(GMC) ratio (Sh_NTHi-Mcat/NTHi-Mcat) is above<br/>a limit of 0.667 for all anti-PD, anti-PE, anti-PilA,<br/>anti-UspA2.</li> </ul> | |

The following modification of the primary objective will be applicable if the per-protocol set is not reached for the Sh NTHi-Mcat 6 group:2

#### Confirmatory

To demonstrate the non-inferiority (NI) of the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 months after Shingrix vaccine versus the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine alone.

#### Criterion:

Lower limit (LL) of the 2-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio (Sh NTHi-Mcat/NTHi-Mcat) is above a limit of 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2

#### Humoral immune response

Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations 1 month after Dose 2 of NTHi-Mcat vaccine in the Sh NTHi-Mcat 3 group (Day 241) and Sh NTHi-Mcat 1 group (Day 181) compared to antibody concentrations 1 month after Dose 2 in the NTHi-Mcat group (Day 91).1

The following modification of the primary objective will be applicable if the per-protocol set is not reached for the Sh NTHi-Mcat 6 and Sh NTHi-Mcat 3 groups:3

To demonstrate the non-inferiority (NI) of the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 month after Shingrix vaccine versus the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine alone.

## Criterion:

Lower limit (LL) of the 2-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio (Sh\_NTHi-Mcat/NTHi-Mcat) is above a limit of 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2.

Humoral immune response

Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations 1 month after Dose 2 of NTHi-Mcat vaccine in the Sh NTHi-Mcat 1 group (Day 181) compared to antibody concentrations 1 month after Dose 2 in the NTHi-Mcat group (Day 91).1

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

| Objectives | Endpoints |
|---|---|
| | condary |
| Descriptive To evaluate the safety and reactogenicity profile of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine or when administered alone. | <ul> <li>Solicited local and general adverse events (AEs) <ul> <li>Occurrence of each solicited local and general adverse event (AE), reported during a 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after Dose 1 and after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine, in all subjects in all groups.</li> </ul> </li> <li>Unsolicited AEs <ul> <li>Occurrence of any unsolicited AEs, reported during a 30-day follow- up period (i.e. day of vaccination and 29 subsequent days) after Dose 1 and after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine, in all subjects in all groups.</li> </ul> </li> <li>Serious AEs <ul> <li>Occurrence of any SAE reported from first vaccination (Day 1) to Day 331 in all subjects in all groups.</li> <li>Occurrence of any SAE, reported from Day 331 to Day 661 in all subjects in all groups.</li> <li>Potential immune-mediate diseases (pIMD)</li></ul></li></ul> |
| To describe the humoral immune response of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine or when administered alone. | <ul> <li>Humoral response <ul> <li>Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations and seropositivity in all subjects before Dose 1 (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group).<sup>1,4</sup></li> </ul> </li> </ul> |
| <u>Descriptive</u> | CMI response |
| To describe the cell mediated immune (CMI) response (CD4+ T-cells) of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine or when NTHi-Mcat is administered alone, in the CMI response sub-cohort. | <ul> <li>NTHi-specific and Mcat-specific CMI responses as measured by flow cytometry ICS (frequency of specific CD4+ T-cells expressing at least 2 different markers among CD40 ligand (CD40L), interleukin (IL)-2, IL-13, IL-17, interferon gamma (IFN-γ), tumour necrosis factor alpha (TNF-α) upon in vitro stimulation) before Dose 1 (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group) in the CMI response sub-cohort.5</li> </ul> |

OL: ...

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

| Objectives | Endpoints |
|---|---|
| Ţ | Tertiary |
| <u>Descriptive</u> | CMI response |
| <ul> <li>To describe the CMI response (CD8+ T-cells) of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after <i>Shingrix</i> vaccine or when NTHi-Mcat is administered alone, in the CMI response subcohort.</li> <li>To explore the T-helper profile of the PD-, PE-, PilA-, UspA2-specific CD4+/ CD8+ T cell responses.</li> </ul> | <ul> <li>NTHi-specific and Mcat-specific CMI responses as measured by flow cytometry ICS (frequency of specific CD8+ T-cells expressing at least 2 different markers among CD40L,IL-2, IL-13, IL-17, IFN-γ, TNF-α upon in vitro stimulation) before Dose 1 (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group) in the CMI response sub-cohort.5</li> </ul> |
| | <ul> <li>T-helper profile <ul> <li>T-helper profile of the specific T-cell response in T-helper 1, T-helper 2 and T-helper 17 based on the specific expression of respectively IFN- γ, IL-13 and IL-17 before Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group) in the CMI subcohort. Frequencies of specific CD4+/CD8+ T cells per 10<sup>6</sup> cells expressing combinations of cytokines/activation markers will be explored.<sup>1</sup></li> </ul> </li> </ul> |

<sup>&</sup>lt;sup>1</sup> Given the different intervals between vaccines, the label for study visits or contacts varies between treatment groups and as such the Visit/contact label varies. Please refer to the study design diagram (Figure 1).

<sup>&</sup>lt;sup>2</sup> A descriptive analysis where the 95% confidence intervals around the geometric mean concentration (GMC) ratio of the Sh\_NTHi-Mcat\_6 group will be presented with all available data. The descriptive analysis may be used to support the interval between Shingrix and NTHi-Mcat vaccines administration

<sup>&</sup>lt;sup>3</sup> A descriptive analysis where the 95% confidence intervals around the geometric mean concentration (GMC) ratio of the Sh\_NTHi-Mcat\_6 and Sh\_NTHi-Mcat\_3 groups will be presented with all available data. The descriptive analysis may be used to support the interval between Shingrix and NTHi-Mcat vaccines administration

<sup>&</sup>lt;sup>4</sup> Cut-off for seropositivity will be the lower limit of quantification (LLOQ) of the assay.

<sup>&</sup>lt;sup>5</sup> Refer to Section 5.3.1 of the study protocol for details regarding the CMI sub-cohort.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 4. ANALYSIS SETS

#### 4.1. Definition

| Analysis Set | Description |
|---|---|
| Enrolled | All subjects who signed informed consent |
| Exposed (ES) | All subjects who received at least 1 dose of the study treatment. The allocation in a group is done in function of the administered treatment. |
| Full analysis (FAS) | All subjects who received at least 1 dose of the study treatment and have post-vaccination immunogenicity data |
| Modified full analysis (mFAS) | All subjects who received full study treatment course to which they are randomized and have post-vaccination immunogenicity data |
| Per protocol (PPS) | All subjects who received full study treatment course to which they are randomized and have post-vaccination data (mFAS) minus subjects with protocol deviations that lead to exclusion |
| Unsolicited safety | All subjects who received at least 1 dose of the study treatment¹ (exposed set) that report unsolicited AEs or that report not having unsolicited AEs |
| Solicited safety | All subjects who received at least 1 dose of the study treatment¹ (exposed set) who have solicited safety data |

<sup>&</sup>lt;sup>1</sup> Study treatment refers to the NTHi-Mcat vaccine. Please refer to Section 4.1.1 for additional details.

#### 4.1.1. Additional considerations

The Enrolled set includes all subjects who signed informed consent, excluding subjects withdrawn prior to randomization (e.g. screening failures).

For the Unsolicited and Solicited safety sets, 1 dose of the study treatment refers to the administration of at least 1 dose of the NTHi-Mcat vaccine, in line with the study analysis of solicited and unsolicited AEs. In addition, subjects exposed to *Shingrix* only (if any) will be included in an extra group named "Shingrix only" for the safety analyses based on the Exposed Set (ES). Refer to Section 9.1.2 for more details about the algorithm to attribute subjects to groups for the purpose of safety analyses.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Details are provided below for each set.

## 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (study vaccine not administered at all), code 800 (fraudulent data) and code 900 (invalid informed consent) will be used for identifying subjects eliminated from the ES.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

Subjects assigned to code 1030.b (not administering any NTHi-Mcat vaccine), but not to code 1030 will be identified as subjects belonging to the "Shingrix only" group.

# 4.2.2. Elimination from Full analysis set (FAS)

## 4.2.2.1. Excluded subjects

A subject will be excluded from the FAS analysis under the following conditions:

| Code | Condition under which the code is used | Visit (V) (timepoints) where the code is applicable | Applicable for endpoint<br>[HUM=humoral<br>response, CMI=CMI<br>response] |
|---|---|---|---|
| 800 | Fraudulent data | All | HUM, CMI |
| 900 | Invalid informed consent | All | HUM, CMI |
| 1030 | Study vaccine not administered at all | All | HUM, CMI |
| 2100.a | Humoral immune response results not available post-vaccination | V6_1, V6_3, V6_6, V4 | HUM |
| 2100.b | CMI response results not available post-vaccination | V6_1, V6_3, V6_6, V4 | CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

Note: in case a subject is bled but blood sample is not planned per study protocol (code 2130), the unexpected sample is eliminated from the analysis, but subject is retained.

## 4.2.3. Elimination from Modified full analysis set (mFAS)

## 4.2.3.1. Excluded subjects

A subject will be excluded from the mFAS analysis <u>if excluded from the FAS</u> and under the following additional conditions:

| Code | Condition under which the code is used | Visit (V) (timepoints) where the code is applicable | Applicable for endpoint<br>[HUM=humoral<br>response, CMI=CMI<br>response] |
|---|---|---|---|
| 1030.b | Not administering any NTHi-Mcat vaccine | All | HUM, CMI |
| 1070.a | Incomplete treatment course | All | HUM, CMI |
| 1070.a | Other deviations related to wrong treatment administered (including randomization failure) | All | HUM, CMI |
| 2080 | Subjects did not comply with Sh_NTHi-<br>Mcat vaccination schedule | V3_1, V3_3, V3_6 | HUM, CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 4.2.4. Elimination from Per-protocol analysis set (PPS)

## 4.2.4.1. Excluded subjects

A subject will be excluded from the PPS analysis <u>if excluded from the mFAS</u> and under the following additional conditions:

| Code | Condition under which the code is used | Visit (V)<br>(timepoints)<br>where the code<br>is applicable | Applicable for endpoint [HUM=humoral response, CMI=CMI response] |
|---|---|---|---|
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol | All | HUM, CMI |
| 1070 | Vaccination not according to protocol | All | HUM, CMI |
| 1080 | Vaccine temperature deviation | All | HUM, CMI |
| 1090 | Expired vaccine administered | All | HUM, CMI |
| 2010 | Protocol violation (inclusion/exclusion criteria) | All | HUM, CMI |
| 2040 | Administration of any medication forbidden by the protocol | All | HUM, CMI |
| 2050 | Medical condition forbidden by the protocol | All | HUM, CMI |
| 2080 | Subjects did not comply with vaccination schedule | All | HUM, CMI |
| 2090.a | Subjects did not comply with blood sample schedule (sample for humoral immune response) | All | HUM |
| 2090.b | Subjects did not comply with blood sample schedule (sample for CMI response) | All | CMI |
| 2100.a | Humoral immune response results not available | All | HUM |
| 2100.b | CMI response results not available | All | CMI |
| 2120.a | Obvious incoherence or abnormality or error in data (data on humoral immune response) | All | HUM |
| 2120.b | Obvious incoherence or abnormality or error in data (data on CMI response) | All | CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort. In case of missed assessment or assessment not properly performed, the codes 2100c and 2120c can be applicable; decision is taken case by case.

## 4.2.5. Elimination from unsolicited and solicited safety set

### 4.2.5.1. Excluded subjects

## 4.2.5.1.1. Unsolicited safety set

Code 1030.b (not administering any NTHi-Mcat vaccine), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1150 (no post-vaccination safety data) will be used to identify subjects eliminated from the unsolicited safety set.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

Code 1150 will be attributed to subjects if <u>all</u> the following conditions are met: subject did not complete the safety assessment following the 7-day follow-up period after NTHi-Mcat vaccinations (i.e. phone contacts), did not return the pDiary, did not return for the scheduled visit 30-days after the NTHi-Mcat vaccinations and did not report any unsolicited AE.

Code 1070.a will be used to identify subjects eliminated from the Unsolicited Safety Set by visit when the NTHi-Mcat vaccination is not administered at that visit.

## 4.2.5.1.2. Solicited safety set

Code 1030.b (not administering any NTHi-Mcat vaccine), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data) will be used to identify subjects eliminated from the solicited safety set.

Code 1070.a will be used to identify subjects eliminated from the Solicited Safety Set by visit when the NTHi-Mcat vaccination is not administered at that visit.

# 5. STATISTICAL ANALYSES

Note that standard data derivation rules and statistical methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and statistical methods will be described in Section 9.

## 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (including age at first study vaccination in years, gender, race, ethnicity and smoking status) will be summarized by study group and overall, using descriptive statistics:

- Frequency tables will be generated for categorical variables such as smoking status.
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age, height and weight.

Withdrawal status will be summarized by group using descriptive statistics:

- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal
- The number of subjects enrolled into the study as well as the number of subjects excluded from the PPS and mFAS will be tabulated.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 5.1.2. Additional considerations

Summaries of demographic/baseline characteristics will include: age, country, centre, gender, race, ethnicity, smoking status, pack-years and vital signs (including body mass index [BMI]).

# 5.2. Exposure

## 5.2.1. Analysis of exposure planned in the protocol

None.

#### 5.2.2. Additional considerations

The number and percentage of subjects who received study vaccine doses will be tabulated for each study group (based on the ES).

# 5.3. Immunogenicity

## 5.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PPS. A supplementary analysis may be based on the mFAS.

| Endpoint | Statistical analysis methods |
|---|---|
| Primary | Between group assessment Considering the sampling timepoint at 1 month after Dose 2 of NTHi-Mcat vaccine, the 2-sided 95% CIs for the group GMC ratio (Sh_NTHi-Mcat_1; _3; _6 group over NTHi-Mcat group) of anti-PD, anti-PE, anti-PilA, anti-UspA2 will be computed using an analysis of covariance (ANCOVA) model on the logarithm10 transformation of the concentrations. The ANCOVA model will include study group, smoking status (current or former), age category (50–59, 60–69, 70–80 years of age) and centre as factors and the antibody concentration before Dose 1 as covariate. |
| | Non-inferiority for a specific time-lag will be claimed if the lower limit of the 2-sided 95% CI for the GMC ratio will be above 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2. The sequential procedure for multiple time-lags will be used: starting from the 6-months lag, the 3-months NI will be tested only if the 6-months NI will be demonstrated, while the 1-month NI will be tested only if the 6-months and 3-months NI will be both demonstrated. |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

| | Statistical Analysis Plan Amendment 2 |
|---|---|
| Endpoint | Statistical analysis methods |
| The following modification of the primary objective will be applicable if the per-protocol set is not reached for the Sh_NTHi-Mcat_6 group:1 | Considering the sampling timepoint at 1 month after Dose 2 of NTHi-Mcat vaccine, the 2-sided 95% CIs for the group GMC ratio (Sh_NTHi-Mcat_1; _3 group over NTHi-Mcat group) of anti-PD, anti-PE, anti-PilA, anti-UspA2 will be computed using an analysis of covariance (ANCOVA) model on the logarithm10 transformation of the concentrations. The ANCOVA model will include study group, smoking status (current or former), age category (50–59, 60–69, 70–80 years of age) and centre as factors and the antibody concentration before Dose 1 as covariate. Non-inferiority for a specific time-lag will be claimed if the lower limit of the 2-sided 95% CI for the GMC ratio will be above 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2. The sequential procedure for multiple time-lags will be used: starting from the 3-months lag, the 1-month NI will be tested only if the 3-months NI will be demonstrated. |
| The following modification of the primary objective will be applicable if the per-protocol set is not reached for the Sh_NTHi-Mcat_6 and the Sh_NTHi-Mcat_3 groups:2 | Considering the sampling timepoint at 1 month after Dose 2 of NTHi-Mcat vaccine, the 2-sided 95% CIs for the group GMC ratio (Sh_NTHi-Mcat_1 group over NTHi-Mcat group) of anti-PD, anti-PE, anti-PilA, anti-UspA2 will be computed using an analysis of covariance (ANCOVA) model on the logarithm10 transformation of the concentrations. The ANCOVA model will include study group, smoking status (current or former), age category (50–59, 60–69, 70–80 years of age) and centre as factors and the antibody concentration before Dose 1 as covariate. Non-inferiority for a specific time-lag will be claimed if the lower limit of the 2-sided 95% CI for the GMC ratio will be above 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2. |
| | Secondary endpoints |
| Secondary - humoral | Within group assessment For each study group, for each sampling timepoint and for each antigen, the following statistics will be computed: Seropositivity rates with exact 95% CI (seropositivity defined using the assay lower limits of quantification [LLOQ]) Adjusted and unadjusted GMCs with 95% CI (adjustment by ANCOVA model, as specified above) The range and distribution of antibody concentrations The distribution of antibody concentrations for each antigen will be displayed using reverse cumulative distribution curves. |
| Secondary –cell-<br>mediated immune<br>response | CMI response induced by the NTHi-Mcat candidate vaccine will be evaluated, presenting the frequencies of antigen-specific CD4+ T cells per 10 <sup>6</sup> cells. The specific CD4+ T cells being identified as the CD4 + T cells expressing at least 2 different markers among CD40 Ligand (CD40L), IL-2, TNF- α, IFN- γ, IL-13 and IL-17 upon in vitro stimulation. Descriptive statistics (Min, Q1, Median, Mean, Q3 & Max) will be reported for each group at pre-Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh-NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group). |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

| Endpoint | Statistical analysis methods |
|---|---|
| Tertiary –cell-<br>mediated immune<br>response | <ul> <li>CMI response induced by the NTHi-Mcat candidate vaccine will be evaluated, presenting the frequencies of antigen-specific CD8+T cells per 10<sup>6</sup> cells. The specific CD8+T cells being identified as the CD8+ T cells expressing at least 2 different markers among CD40L, IL-2, TNF- α, IFN- γ, IL-13 and IL-17 upon in vitro stimulation.</li> <li>CMI response as the frequencies of specific CD4+/CD8+ T cells per 10<sup>6</sup> cells expressing any combination of cytokines/activation markers will be determined. The T-helper profile of the specific T-cell response in T-helper 1, T-helper 2 and T-helper 17 based on the specific expression of respectively IFN-γ, IL-13 and IL-17 will be characterized.</li> <li>Descriptive statistics (Min, Q1, Median, Mean, Q3 &amp; Max) will be reported for each group at pre-Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh-NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group).</li> </ul> |

<sup>&</sup>lt;sup>1</sup> A descriptive analysis where the 95% confidence intervals around the geometric mean concentration (GMC) ratio of the Sh\_NTHi-Mcat\_6 group will be presented with all available data. The descriptive analysis may be used to support the interval between Shingrix and NTHi-Mcat vaccines administration

#### 5.3.2. Additional considerations

The supplementary analysis based on the mFAS will be performed if the percentage of mFAS subjects excluded from the PPS is more than 10%.

### 5.3.2.1. Analysis of humoral response

#### Hypothesis related to the primary objective

The global null hypothesis related to the primary objective of the study is that at least 1 GMC ratio (Sh\_NTHi-Mcat over NTHi-Mcat) among anti-PD, anti-PE, anti-PilA, anti-UspA2 is inferior or equal to 0.667 in all time-lags under investigation at 1 month post-Dose 2 of NTHi-Mcat vaccine. This must be rejected in favour of the alternative hypothesis that all 4 GMCs (anti-PD, anti-PE, anti-PilA, anti-UspA2) are non-inferior in at least one time-lag group. Family-wise type I error is fixed at 2.5% (1-sided).

#### Geometric mean concentration and geometric mean concentration ratio

For each antigen and study group, at 1 month after Dose 2 of NTHi-Mcat vaccine, adjusted GMCs and GMCs ratios with corresponding 95% CIs will be obtained exponentiating (base 10) the least square means and the lower and upper limits of the 95% CIs derived from the ANCOVA model. The ANCOVA model will be implemented in SAS, similarly to the following code:

```
PROC GLM data=<dataset>;
BY antigen;
class group age smoking_status centre;
MODEL log(concentr) = group age smoking_status centre log(pre_concentr);
LSMEAN group / CL PDIFF ALPHA=0.05;
RUN;
```

<sup>&</sup>lt;sup>2</sup> A descriptive analysis where the 95% confidence intervals around the geometric mean concentration (GMC) ratio of the Sh\_NTHi-Mcat\_6 and Sh\_NTHi-Mcat\_3 groups will be presented with all available data. The descriptive analysis may be used to support the interval between Shingrix and NTHi-Mcat vaccines administration

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

Contrasts to be included: Sh\_NTHi-Mcat\_6 vs NTHi-Mcat, Sh\_NTHi-Mcat\_3 vs NTHi-Mcat, Sh\_NTHi-Mcat\_1 vs NTHi-Mcat.

In addition, unadjusted GMCs and GMRs will be presented for each timepoint (pre-Dose 1 and post-Dose 2 of NTHi-Mcat vaccine) with a descriptive purpose.

## Permutation test (sensitivity analysis on primary objectives)

Based on the covariate-adaptive treatment assignment algorithm (see Section 10.3), the following permutation test will be performed as a sensitivity analysis on the primary objectives<sup>1</sup> [Wiens, 2006, Hasegawa, 2009 and Ernst, 2004] in the PPS.

For each antigen, let  $\mathbf{X}$ =( $X_1$ , ...,  $X_N$ ) the logarithmically-transformed antibody concentrations for the NTHi-Mcat group and  $\mathbf{Y}_{1/3/6}$ =( $Y_1$ , ...,  $Y_N$ ) the logarithmically-transformed antibody concentrations for one of the Sh\_NTHi-Mcat groups at 1 month after Dose 2 of NTHi-Mcat vaccine, a non-inferiority permutation test can be obtained from a superiority permutation test on  $\dot{\mathbf{X}}$ =( $X_1$ , ...,  $X_N$ ) against  $\dot{\mathbf{Y}}_{1/3/6}$ =( $X_1$ ) with  $X_1$ 0 = -log<sub>10</sub>(0.667).

The original treatment assignment algorithm will be used to re-randomize subjects while keeping antibody concentrations, covariates and entry order as observed. The procedure will be as follows:

- 1. Fit the ANCOVA model to obtain the test statistics  $T*_{1/3/6}$  for the superiority of  $\dot{\mathbf{X}}$  against  $\dot{\mathbf{Y}}_{1/3/6}$ .
- 2. Estimate the distribution of the test statistics with R=10000 repetitions of the following 2 steps:
  - a. Re-randomize treatment assignment of all 4 groups (original algorithm).
  - b. Re-fit the ANCOVA model to re-obtain the test statistics  $T_{1/3/6}$ .
- 3. Derive the permutation p-values associated to the observed test statistics (from step 1) based on the empirical distributions in Step 2

$$\mathbf{p}_{1/3/6} = \mathbf{M} + 1/\mathbf{R} + 1$$

Where M is the number of repetitions such that  $T_{1/3/6} \ge T^*_{1/3/6}$ .

<sup>&</sup>lt;sup>1</sup> if the primary objective, following the assessment in term of number of subjects in PPS, is based on a reduce number of groups, the permutation p-values associated to the observed test statistics will be derived only for the groups participating to the primary objective.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

### Seropositivity rate and fold increase

For each antigen, timepoint and study group, the seropositivity rate (defined as the proportion of subjects with an antibody concentration greater or equal to the assay cutoff) with exact 95% CIs will be computed using the method referenced in section 10.1.5.1. Assay cut-offs are reported in section 9.1.1. In addition, percentages of subjects with a 2/4/8-fold increase will be presented with associated 95% CI.

## **Reverse cumulative distribution curves**

Reverse cumulative distribution (RCD) curves for antibody concentrations will be plotted: the x-axis represents the antibody concentrations value (log-10 scale), while the y-axis the percentage of subjects having a log-transformed antibody value greater or equal to the corresponding x-value.

## 5.3.2.2. Analysis of CMI response

The frequency of **antigen-specific** CD4+ or CD8+ T-cells for each individual subject is calculated as the difference between the frequency of CD4+ or CD8+ T-cells producing at least 2 activation markers among CD40 Ligand (CD40L), IL-2, TNF-  $\alpha$ , IFN-  $\gamma$ , IL-13 and IL-17, upon *in vitro* stimulation with the antigen (induction condition) minus the frequency of CD4+ or CD8+ T-cells producing at least 2 activation markers upon in vitro stimulation in medium only (background condition). For descriptive statistics purposes, differences less or equal to zero (0) are imputed to 1.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

# 5.4. Analysis of safety and reactogenicity

# 5.4.1. Analysis of safety and reactogenicity planned in the protocol

All safety analyses will be performed on the solicited safety set, unsolicited safety set and exposed set.

| Endpoint | Statistical analysis methods |
|---|---|
| Secondary | Within group assessment The percentage of subjects with at least 1 local adverse event (AE) (solicited and unsolicited), with at least 1 general AE (solicited and unsolicited) and with any AE during the 7-days solicited follow-up period and the 30-days follow-up period will be tabulated by group with exact 95% CI after each NTHi-Mcat vaccine dose and overall. The percentage of NTHi-Mcat doses followed by at least 1 local AE (solicited and unsolicited), by at least 1 general AE (solicited and unsolicited) and by any AE will be tabulated by group with exact 95% CI. The same calculations will be performed for AEs rated as Grade 3, for AEs causally related to vaccination and Grade 3 AEs causally related to vaccination. The percentage of subjects reporting each individual solicited local and general AE during the 7-days solicited follow-up period after each dose of NTHi-Mcat vaccine will be tabulated by group with exact 95% CI. The percentage of NTHi-Mcat doses followed by each individual solicited local and general AE will be tabulated by group with exact 95% CI. Fever will be reported per 0.5°C cumulative increments. For all solicited symptoms, the same tabulation will be performed for Grade 3 AEs. |
| | The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) Dictionary for Adverse Event Terminology. The percentage of subjects with at least 1 report of unsolicited adverse event classified by the MedDRA and reported up to 30 days after NTHi-Mcat vaccinations will be tabulated by group with exact 95% CI. The same tabulation will be performed for Grade 3 unsolicited adverse events, for unsolicited adverse events with a causal relationship to vaccination and for Grade 3 AEs causally related to vaccination. The number of subjects who experienced any serious adverse event (SAE) or any potential |
| | immune-mediated disease (pIMD) from Day 1 to Day 331 and from Day 331 to Day 661 will be reported. |
| | The number of subjects who experienced any AE leading to study withdrawal, from first vaccination up to study conclusion, or any SAE related to study participation or concurrent GSK medication/vaccination, during the entire study period, will be reported. |
| | A summary of subjects reporting concomitant medication/product will be provided. |

## 5.4.2. Additional considerations

## 5.4.2.1. Analysis of solicited AEs

The analysis of solicited AEs will be performed on the Solicited safety set.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals as follows:

Grade 0: <20 mm diameter

Grade 1:  $\geq$ 20 mm to  $\leq$ 50 mm diameter Grade 2:  $\geq$ 50 mm to  $\leq$ 100 mm diameter

Grade 3: >100 mm diameter

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

Temperature (i.e. fever) will be scored at GSK Biologicals as follows:

Grade 0: <37.5°C

Grade 1: 37.5°C to 37.9°C Grade 2: 38.0°C to 38.9°C

Grade 3: >39.0°C

Fever, defined as a body temperature of  $\geq$ 37.5°C irrespective of route of measurement, will be integrated to the summaries as a general AE.

In addition, body temperature will be broken down into 0.5°C increments:

- < <36.0
- 36.0 36.4
- 36.5 36.9
- 37.0 37.4
- 37.5 37.9
- 38.0 38.4
- 38.5 38.9
- 39.0 39.4
- 39.5 39.9
- >40.0

Compliance of subjects in completing solicited AEs information will be reported as the percentage of subjects completing at least 80% of the diary entries related to local and general solicited AEs.

#### 5.4.2.2. Analysis of unsolicited AEs

The analysis of unsolicited AEs will be performed on the Unsolicited safety set.

Analysis of unsolicited AEs will be also stratified on AEs with a causal relationship to NTHi-Mcat vaccination.

#### 5.4.2.3. Combined analysis of solicited and unsolicited AEs

The combined analysis of solicited and unsolicited AEs will be performed on the Unsolicited safety set.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

Solicited AEs will be coded by MedDRA as per the following codes:

| Solicited symptom | Preferred Term code | Corresponding Preferred Term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Redness | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Gastrointestinal symptoms | 10017944 | Gastrointestinal disorder |
| Myalgia | 10028411 | Myalgia |
| Chills | 10008531 | Chills |
| Fever | 10037660 | Pyrexia |

Combined analysis of solicited and unsolicited AEs will be also stratified on AEs with a causal relationship to NTHi-Mcat vaccination (all solicited AEs are considered causally related).

### 5.4.2.4. Analysis of SAEs and pIMDs

The analysis of SAEs and pIMDs will be performed on the Exposed Set (ES).

Analysis of SAEs will include:

- All SAEs from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
- Fatal SAEs from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
- Related SAEs:
  - To any study vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
  - To the NTHi-Mcat vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661, from the day of the first NTHi-Mcat vaccination up to 1 month following the second dose, from the day of the first NTHi-Mcat vaccination up to 6 months following the second dose and from the day of the first NTHi-Mcat vaccination up to 12 months following the second dose (all groups except "Shingrix only").
  - To Shingrix vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661 (all groups except NTHi-Mcat).

Analysis of pIMDs will include all occurrences from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 5.4.2.5. Other safety analyses

Medications will be coded using GSKDRUG dictionary.

All collected concomitant medications and vaccinations will be listed. In addition, prior and concomitant vaccinations will be summarized. In case of pregnancies during the study, follow-up data and pregnancy outcomes will be described in detail.

## 6. ANALYSIS INTERPRETATION

Except for analysis on primary objectives, with predefined success criteria and an appropriate type I error control, comparative analyses are descriptive with the aim to characterize the difference between groups.

With respect to confirmatory analyses on primary objectives the interpretation will be done in a hierarchical manner, except if only the group Sh\_NTHi-Mcat\_1 reached the number of subjects planned in the PPS, in this case we will have only one comparison to interpret.

In case of sequential testing will be applied, each non inferiority can only be concluded if all the associated criteria are met and all previous non inferiority have been concluded (see Figure 2): starting from the 6-months lag, the 3-months NI can be achieved only if the 6-months NI is demonstrated, while the 1-month NI can be achieved only if the 6-months and 3-months NI are both demonstrated. Starting from the 3-months lag, the 1-month NI can be achieved only if the 3-months NI is demonstrated.

This sequential procedure enables to control the overall type I error below 2.5% (one-sided) [Dmitrienko, 2009].

Figure 2 Sequence for evaluating the primary objective in order to control the overall type I error below 2.5% (one-sided) in case all groups reached the number of subjects planned in the PPS



209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

If the per-protocol sample size is not reached in the Sh\_NTHi-Mcat\_6 group, the sequential procedure enables to control the overall type I error below 2.5% (one-sided) [Dmitrienko, 2009] will be:



## 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

The integrated clinical study report (CSR) will contain at least the final analyses of all primary and secondary endpoints. If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These analyses will be documented in annex(es) to the study report.

The analyses will be performed stepwise:

- A final analysis of immunogenicity, safety and reactogenicity for all subjects up to and including Day 331 ('Epoch 001') will be performed in a first step.
  - A complete study report containing all data of 'Epoch 001' will be written and made available to the investigators at this stage.
- Analysis conducted on the data collected for all subjects from Day 331 up to and including Day 661 ('Epoch 002') will be performed in a second step.

An integrated CSR containing all data from Epoch 001 and Epoch 002 will be written and made available to the investigators.

| Description | Disclosure Purpose<br>(CTRS=public posting, SR=study report, internal) |
|---|---|
| Final Analysis Epoch 001 | Web disclosure (CTRS), Study report (SR) |
| Analysis of Follow-up Epoch | Web disclosure (CTRS), Study report (SR) |

# 7.2. Statistical considerations for interim analyses

No interim analysis is planned for this study. Data up to and including Day 331 are considered 'final' and completed data, while the remaining safety data are considered long-term safety follow-up.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 8. CHANGES FROM PLANNED ANALYSES

Not applicable

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in Section 10.1

#### 9.1. Data derivation

## 9.1.1. Assay cut-offs for serology results

| Component | Method | Unit <sup>1</sup> | Assay cut-off¹ |
|-------------------------|--------|-------------------|----------------|
| anti-PD antibody | ELISA | EU/mL | 153 |
| anti-PE antibody | ELISA | EU/mL | 25 |
| anti-PilA antibody | ELISA | EU/mL | 16 |
| anti-UspA2 IgG antibody | ELISA | EU/mL | 38 |

ELISA = Enzyme Linked Immunosorbent Assay; EU/ml = ELISA unit per millilitre; Ig = immunoglobulin; PD = protein D; from NTHi; PE = protein E from NTHi; PilA = type IV pili subunit from NTHi; UspA2 = ubiquitous surface protein A2 from Mcat

## 9.1.2. Attributing subjects to time-lag groups

For the purpose of safety analyses, the following rule will be used to attribute exposed subjects to a specific group.

- If a subject receives no *Shingrix* vaccination → NTHi-Mcat group
- If a subject receives at least 1 *Shingrix* vaccination, but no NTHi-Mcat vaccination → "Shingrix only" group
- If a subject receives at least 1 *Shingrix* vaccination and at least 1 NTHi-Mcat vaccination, the difference, in days, between the latest Shingrix vaccination and the earliest NTHi-Mcat vaccination will be computed and converted in months (diff):
  - diff ≤ 2  $\rightarrow$  Sh\_NTHi-Mcat\_1 group
  - 2 < diff ≤ 4.5  $\rightarrow$  Sh\_NTHi-Mcat\_3 group
  - diff > 4.5  $\rightarrow$  Sh NTHi-Mcat 6 group

#### 9.2. Statistical Method

Not applicable

<sup>1</sup> Assay cut-off and unit might be subject to change during the course of the study (e.g. in case of assay reoptimization, qualification, (re)validation or standardization). In this case, this will be documented in the clinical study report.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in Section 9 (additional study-specific rules).

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the eCRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one

## 10.1.2. Handling of missing data

## 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30th.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

## 10.1.2.3. Daily recording of solicited symptoms

#### 10.1.2.3.1. Studies with paper diaries

Denominators for the summary of local (or general) solicited symptoms will be calculated using the number of subjects who respond "Yes" or "No" to the question concerning the occurrence of local (or general) symptoms.

When a specific symptom is marked as having not occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=N for the specified post-vaccination period for the symptom in question), all daily measurements will be imputed as Grade 0.

When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

When the occurrence of a specific symptom is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-vaccination period for the symptom in question) but the group of symptoms (local or general) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

The following table shows how subjects contribute to each category for a specific solicited symptom over the Day X to Day Y post-vaccination period:

| Solicited symptom category | Subjects included in the calculation of the numerator |
|---|---|
| Any | All subjects with at least one occurrence of the symptom at Grade 1, Grade 2, or Grade 3 between Day X and Day Y or with the symptom marked as present and at least one missing daily recording between Day X and Day Y |
| At least Grade 1 | All subjects with at least one occurrence of the symptom at Grade 1, Grade 2, or Grade 3 between Day X and Day Y |
| At least Grade 2 | All subjects with at least one occurrence of the symptom at Grade 2 or Grade 3 between Day X and Day Y |
| At least Grade 3 | All subjects with at least one occurrence of the symptom at Grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### 10.1.3. Data derivation

## 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

## 10.1.3.2. Body mass index (BMI)

BMI will be calculated as follows:

 $BMI = (weight in kilograms) / (height in meters)^2$ 

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

## 10.1.3.4. Geometric mean concentrations (GMCs)

GMC calculations are performed by taking the inverse logarithm of the mean of the log-10 concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

## 10.1.3.5. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus 1 day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the consecutive days with the symptom reported at Grade 1 or higher. The duration of solicited events at a specific grade (e.g. Grade 3) will be calculated as the sum of the consecutive days with the symptom reported at that grade. The same rule applies for solicited events ongoing at the end of the solicited follow-up period considering the maximum intensity reported.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event eCRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

## 10.1.3.8. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarised, each event recorded as having occurred during a specific period will be counted as the number of occurrences the event is consecutively reported (at Grade 1 or higher). When the occurrences of solicited adverse events at a specific grade are summarised, each event recorded as having occurred at that grade during a specific period will be counted as the number of occurrences the event is consecutively reported at that grade.

## 10.1.4. Display of decimals

## 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

## 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with 1 more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with 1 decimal will be displayed with 2 decimals.

### 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, BMI, pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values

The maxima and minima of transformed height variables will be displayed with no decimals.

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values below 10kg where 1 decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with 1 decimal.

## 10.1.4.4. Serological summary statistics

The number of decimals used when displaying GMCs and their confidence limits is shown in the following table:

| GMC value | Number of decimals to display |
|----------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the 1 with the higher number of decimals). For example, if GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 10.1.5. Statistical methodology

## 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Mietinnen and Nurminen [Miettinen, 1985].

## 10.1.5.3. Adjusted GMC ratios

When between-group GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure.

#### 10.2. TFL ToC

The list of tables, figures and listings (TFL ToC) planned for this study can be found in eTMF folder section 11.1.1.

# 10.3. Randomization method and minimization algorithm

The minimization algorithm used at the GSK internet randomization system (i.e. SBIR) for study NTHI MCAT-009 is based on the following reference: "White SJ, Freedman LS. Allocation of patients to treatment groups in a controlled clinical study. Br J Cancer 1978; 37: 849-857" [White, 1978] and it is described below:

#### **Notations**

- K=3 input values [Centre, Smoking status and Age category] to be used for minimization, each with a weight  $w_k=1$  (k=1,...,K) &  $l_k$  variants.
- I=4 treatment groups [NTHi-Mcat, Sh\_NTHi-Mcat\_6, Sh\_NTHi-Mcat\_3, Sh\_NTHi-Mcat\_1] with randomization ratio a<sub>1</sub>,...,a<sub>I</sub> [1:1:1:1]

#### Algorithm

For a new subject with input value variants  $s_1...s_K$ 

## Step 1: Minimization computation

Step 1.1: Initialize Problem flag to 0

For each input value variant  $s_k$ , compute the number of subjects already enrolled in each treatment group.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

Let  $b_{ik}$  the number for treatment i & input value variant  $s_k$ :  $b_{ik}$  is the total number of subjects already randomized in treatment i and with variant  $s_k$ .

Step 1.2: For each treatment i: compute  $A_i = 1/a_i * sum_k(w_k * b_{ik})$ 

Step 2: determine whether the algorithm is random or deterministic:

Generate R, a random number within [0-1], uniform distribution

Step 3: check determinism

If R < 0.9, go to step 4 (determinism) else go to step 5 (random)

Step 4: determinism

4.1: Identify all treatments with the lowest value A<sub>i</sub>

4.2: Select randomly one of the treatments identified in step 4.1, let it be T.

Go to step 6, if no more treatment then randomization failed

Step 5: randomization

Select randomly one of the treatments, let it be T.

Go to step 6, if no more treatment then randomization failed.

Step 6: treatment allocation

Assign one of the treatment nr. related to treatment T in the subject's center.

If no treatment nr. related to treatment T is available in the subject's center, then go & repeat step 4 (determinism) or 5 (random) while dropping treatment T (set problem flag=1).
209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 2

## 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934; 26:404-13.

Dmitrienko, A., Tamhane, A. C., & Bretz, F. (2009). Multiple testing problems in pharmaceutical statistics. CRC press.

Ernst MD, Permutation Methods: A Basis for Exact Inference. *Statistical Science*, 2004; 19: 676-685.

Hasegawa T, Tango T. Permutation test Following Covariate-Adaptive Randomization in Randomized Controlled Trials. *Journal of Biopharmaceutical Statistics*, 2009; 19: 106-119.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. *Statistics in Medicine*, 1985;4:213-226.

White SJ, Freedman LS. Allocation of patients to treatment groups in a controlled clinical study. *Br J Cancer*, 1978;37: 849-857

Wiens BL, Randomization as basis for inference in noninferiority trials. *Pharmaceutical Statistics*, 2006; 5: 265-271

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | Immunogenicity and safety study of GSK's investigational vaccine (GSK3277511A) when administered in healthy smokers and ex-smokers following receipt of <i>Shingrix</i> vaccine. |
| eTrack study number and<br>Abbreviated Title | 209538 (NTHI MCAT-009) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Amendment 1 Final: 30 January 2020 |

APP 9000058193 Statistical Analysis Plan Template V4 (Effective date: 3June2019)

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | T OF A | BBREVIA | TIONS | | 6 |
| 1. | DOCL | JMENT HI | STORY | | 8 |
| 2. | STUD | Y DESIGN | ١ | | 9 |
| 3. | OBJE | CTIVES A | ND ENDP | OINTS | 11 |
| 4 | A N I A I . | VOIC OFT | | | 40 |
| 4. | 4.1. | | | | |
| | 4.1. | 4.1.1. | | considerations | |
| | 4.2. | | | ing data from Analysis Sets | |
| | | 4.2.1. | Eliminatio | n from Exposed Set (ES) | 13 |
| | | 4.2.2. | Eliminatio | n from Full analysis set (FAS) | 14 |
| | | | 4.2.2.1. | Excluded subjects | 14 |
| | | 4.2.3. | Eliminatio | n from Modified full analysis set (mFAS) | |
| | | | 4.2.3.1. | | 14 |
| | | 4.2.4. | | n from Per-protocol analysis set (PPS) | |
| | | | 4.2.4.1. | Excluded subjects | 15 |
| | | 4.2.5. | | n from unsolicited and solicited safety set | |
| | | | 4.2.5.1. | Excluded subjects | |
| | | | | 4.2.5.1.1. Unsolicited safety set | |
| | | | | 4.2.5.1.2. Solicited safety set | 10 |
| 5. | STAT | ISTICAL A | NALYSES | | 16 |
| | 5.1. | Demogra | aphy | | 16 |
| | | 5.1.1. | | of demographics/baseline characteristics planned | |
| | | <b>5</b> 40 | | tocol | |
| | <b>5</b> 0 | 5.1.2. | | considerations | |
| | 5.2. | 5.2.1. | | of averaging planned in the protocol | |
| | | 5.2.1.<br>5.2.2. | | of exposure planned in the protocol | |
| | 5.3. | | | CONSIDERATIONS | |
| | 5.5. | 5.3.1. | | of immunogenicity planned in the protocol | |
| | | 5.3.2. | | l considerations | |
| | | 0.0.2. | 5.3.2.1. | Analysis of humoral response | |
| | | | 5.3.2.2. | Analysis of CMI response | |
| | 5.4. | Analysis | | and reactogenicity | |
| | | 5.4.1 <sup>°</sup> . | Analysis o | of safety and reactogenicity planned in the | |
| | | 5.4.2. | | considerations | |
| | | | | Analysis of solicited AEs | |
| | | | 5.4.2.2. | , | 22 |
| | | | 5.4.2.3. | Combined analysis of solicited and unsolicited | 00 |
| | | | E 4 O 4 | Applyais of SAEs and pIMDs | 22 |
| | | | 5.4.2.4.<br>5.4.2.5. | Analysis of SAEs and pIMDs | |
| | | | 5.4.2.5. | Other safety analyses | 23 |
| 6. | ANAL | YSIS INTE | ERPRETAT | ΓΙΟΝ | 23 |

| | | | | 209538 (NTHI MCA<br>Statistical Analysis Plan Amend | |
|---|---|---|---|---|---|
| 7. | COND | UCT OF A | ANAI YSES | S | |
| ٠. | 7.1. | | | es | |
| | 7.2. | | | ations for interim analyses | |
| | | | | , | |
| 8. | CHAN | GES FRO | M PLANNI | ED ANALYSES | 25 |
| 9. | NON-S | STANDAR | RD DATA D | ERIVATION RULES AND STATISTICAL | |
| | METH | ODS | | | 25 |
| | 9.1. | Data der | | | |
| | | 9.1.1. | | -offs for serology results | |
| | 0.0 | 9.1.2. | | subjects to time-lag groups | |
| | 9.2. | Statistica | al Method | | 25 |
| 10. | ANNE | | | | |
| | 10.1. | | | tandard data derivations and statistical methods | |
| | | | | events to vaccine doses | |
| | | 10.1.2. | | of missing data | |
| | | | | Dates | |
| | | | | Laboratory data | |
| | | | 10.1.2.3. | , | |
| | | | 10.1.2.4. | 10.1.2.3.1. Studies with paper diaries Unsolicited adverse events | 21<br>28 |
| | | 10.1.3. | - | ration | |
| | | 10.1.0. | 10.1.3.1. | Age at vaccination in years | |
| | | | 10.1.3.2. | Body mass index (BMI) | |
| | | | 10.1.3.3. | Numerical serology results | |
| | | | 10.1.3.4. | Geometric mean concentrations (GMCs) | |
| | | | 10.1.3.5. | Onset day | |
| | | | 10.1.3.6. | Duration of events | 29 |
| | | | 10.1.3.7. | Counting rules for combining solicited and | |
| | | | | unsolicited adverse events | 30 |
| | | | 10.1.3.8. | Counting rules for occurrences of solicited | 00 |
| | | 10 1 1 | Diaplay of | adverse events | |
| | | 10.1.4. | 10.1.4.1. | decimals | |
| | | | 10.1.4.1. | Percentages | |
| | | | 10.1.4.2. | Differences in percentages Demographic/baseline characteristics statistics | 31<br>31 |
| | | | 10.1.4.3. | Serological summary statistics | |
| | | 10.1.5. | | methodology | |
| | | 10.1.5. | 10.1.5.1. | • | |
| | | | 10.1.5.1. | Standardized asymptotic confidence intervals | 02 |
| | | | | around differences in proportions | 32 |
| | | | 10.1.5.3. | | |
| | 10.2. | | | | 32 |
| | 10.3. | Random | ization met | hod and minimization algorithm | 32 |
| 11 | DEEE | DENICES | | | 24 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

# **LIST OF TABLES**

| | | PAGE |
|---------|----------------------------------------------------------|------|
| Table 1 | Study groups, treatment and epochs foreseen in the study | 10 |

4

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

# **LIST OF FIGURES**

| | PA | GE |
|---|---|---|
| Figure 1 | Study design overview | 9 |
| Figure 2 | Sequence for evaluating the primary objective in order to control the overall type I error below 2.5% (one-sided) | 24 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## LIST OF ABBREVIATIONS

AE Adverse event

ANCOVA Analysis of Covariance

ANOVA Analysis of Variance

CI Confidence Interval

CMI Cell-Mediated Immune

eCRF Electronic Case Report Form

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

EU/mL ELISA unit per milliliter

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set

eTMF Electronic Trial Master File

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMR Geometric mean ratio

GSK GlaxoSmithKline

LL Lower Limit

LLOQ Lower Limit of Quantification

MedDRA Medical Dictionary for Regulatory Activities

mFAS Modified Full Analysis Set

NA Not Applicable

NI Non-Inferiority

PD Protocol Deviation

PPS Per-Protocol Set

# 209538 | Statistical Analysis Plan Amendment 1 30 Jan 2020 | TMF-1618943 | 2.0

### CONFIDENTIAL

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

RCD Reverse cumulative distribution

SAE Serious adverse event

SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SDTM Study Data Tabulation Model

SR Study Report

TFL Tables Figures and Listings

ToC Table of Content

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 01 APR 2019 | First version | Protocol Administrative<br>Change 1: 14 DEC<br>2018 |
| 30 JAN 2020 | Amendment 1: Section 5.3.2.1: update to the permutation test algorithm (recommendation from Center for Biologics Evaluation and Research) | Protocol Administrative<br>Change 1: 14 DEC<br>2018 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## 2. STUDY DESIGN

Figure 1 Study design overview



BS C = blood sample for cell-mediated immune response; BS H = blood sample for humoral immune responses/assay development from all subjects; C= Call; D = Day; mth(s) = month(s); NA = not applicable; NM = NTHi-Mcat vaccination; RAND = randomization; S = Safety; Sh = *Shingrix* vaccination; V = Visit Notes:

- <sup>1.</sup> Groups: Sh\_NTHi-Mcat\_1 (NTHi-Mcat vaccine administered 1 month after *Shingrix* vaccine)
- <sup>2</sup> Groups: Sh\_NTHi-Mcat\_3 (NTHi-Mcat vaccine administered 3 months after *Shingrix* vaccine)
- <sup>3.</sup> Groups: Sh NTHi-Mcat 6 (NTHi-Mcat vaccine administered 6 months after *Shingrix* vaccine)
- <sup>4</sup> Patients randomized to the NTHi-Mcat control group will receive the first NTHi-Mcat vaccination at Visit 1 (Day 1) and the second NTHi-Mcat vaccination at Visit 3 (Day 61)
- <sup>5</sup> Blood sample for cell-mediated immune response will be taken from approximately 60 subjects ( ~15 subjects in each group. Refer to Section 5.3.1 of the study protocol for details of the CMI sub-cohort
- <sup>6.</sup> Solicited local and general adverse events reported during a 7-day follow-up period after Dose 1 and after Dose 2 of NTHi-Mcat vaccine, and unsolicited adverse events reported during a 30-day follow-up period after Dose 1 and after Dose 2 of NTHi-Mcat vaccine will be collected
- 7. Safety follow-up

30-JAN-2020 9

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

- **Primary completion date (PCD):** PCD will be 1 month post-Dose 2 of the NTHi-Mcat investigational vaccine (Day 331, based on Sh\_NTHi-Mcat\_6 treatment group).
- End of Study (EoS): Last subject last visit (Day 661).
- **Study groups:** Approximately 540 eligible subjects who will be randomly assigned to 4 study groups in a (1: 1: 1) ratio (Table 1). Please refer to Section 10.1 of the protocol for details related to the determination of sample size.

Table 1 Study groups, treatment and epochs foreseen in the study

| Study Groups | Number Age | | Treatment name | Epochs<br>(Blinding) | |
|---|---|---|---|---|---|
| Study Groups | subjects | (Min-Max) | Treatment name | Epoch 001<br>(open-label) | Epoch 002<br>(open-label) |
| Sh_NTHi-Mcat_1 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| Sh_NTHi-Mcat_3 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| Sh_NTHi-Mcat_6 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| NTHi-Mcat | 135 | 50 – 80 years | NTHi-Mcat | • | • |

- Treatment allocation: Subjects will be allocated to a study group using an automated, electronic System Built for Internet Randomization (SBIR). The randomization algorithm will use a minimization procedure accounting for age category (50–59, 60–69, 70–80 years of age), smoking status (current or former smoker), and centre. Minimization factors will have equal weight in the minimization algorithm.
- **Blinding:** open-label.
- **Data collection:** Electronic Case Report Form (eCRF). Telephone contact. Solicited and unsolicited symptoms will be collected using a subject Diary (paper diary [pDiary]).
- Safety monitoring: Subjects will be observed for at least 60 minutes after each NTHi-Mcat vaccination for any immediate reactions. Solicited local and general AEs occurring during a 7-day follow-up period after each NTHi-Mcat vaccination (i.e. the day of vaccination and the 6 subsequent days) and unsolicited AEs occurring during a 30-day follow-up period after each NTHi-Mcat vaccination (i.e. the day of vaccination and the 29 subsequent days), will be reported via diary cards. In addition, subjects will be asked at Phone contacts if there were any safety concerns in the 7-day follow-up period after each NTHi-Mcat vaccination; this information will be recorded via the appropriate section of the eCRF. Finally, safety assessments will be performed during each clinic visit and safety follow-up calls to collect information on AEs leading to withdrawal, serious adverse events (SAEs), SAEs related to study participation or to a concurrent GSK medication/vaccine, pregnancies, potential immune-mediated diseases (pIMDs), throughout the whole study period.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

# 3. OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Р | rimary |
| <ul> <li>Confirmatory</li> <li>To demonstrate the non-inferiority (NI) of the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine versus the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine alone.</li> <li>Criterion:</li> <li>Lower limit (LL) of the 2-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio (Sh_NTHi-Mcat/NTHi-Mcat) is above a limit of 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2.</li> </ul> | <ul> <li>Humoral immune response</li> <li>Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations 1 month after Dose 2 of NTHi-Mcat vaccine in the Sh_NTHi-Mcat groups (Day 181; Day 241; Day 331) compared to antibody concentrations 1 month after Dose 2 in the NTHi-Mcat group (Day 91).1</li> </ul> |
| · | condary |
| Descriptive To evaluate the safety and reactogenicity profile of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine or when administered alone. | <ul> <li>Solicited local and general adverse events (AEs) <ul> <li>Occurrence of each solicited local and general adverse event (AE), reported during a 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after Dose 1 and after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine, in all subjects in all groups.</li> </ul> </li> <li>Unsolicited AEs <ul> <li>Occurrence of any unsolicited AEs, reported during a 30-day follow- up period (i.e. day of vaccination and 29 subsequent days) after Dose 1 and after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine, in all subjects in all groups.</li> <li>Serious AEs <ul> <li>Occurrence of any SAE reported from first vaccination (Day 1) to Day 331 in all subjects in all groups.</li> <li>Occurrence of any SAE, reported from Day 331 to Day 661 in all subjects in all groups.</li> <li>Potential immune-mediate diseases (pIMD)</li></ul></li></ul></li></ul> |

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

| | Statistical Analysis Plan Amendment 1 |
|---|---|
| Objectives | Endpoints |
| To describe the humoral immune response of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after <i>Shingrix</i> vaccine or when administered alone. | <ul> <li>Humoral response</li> <li>Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations and seropositivity in all subjects before Dose 1 (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group).<sup>1,2</sup></li> </ul> |
| To describe the cell mediated immune (CMI) response (CD4+ T-cells) of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after <i>Shingrix</i> vaccine or when NTHi-Mcat is administered alone, in the CMI response sub-cohort. | <ul> <li>CMI response</li> <li>NTHi-specific and Mcat-specific CMI responses as measured by flow cytometry ICS (frequency of specific CD4+ T-cells expressing at least 2 different markers among CD40 ligand (CD40L), interleukin (IL)-2, IL-13, IL-17, interferon gamma (IFN-γ), tumour necrosis factor alpha (TNF-α) upon in vitro stimulation) before Dose 1 (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group) in the CMI response sub-cohort.1</li> </ul> |
| T | ertiary |
| Descriptive To describe the CMI response (CD8+ T-cells) of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine or when NTHi-Mcat is administered alone, in the CMI response subcohort. To explore the T-helper profile of the PD-, PE-, PilA-, UspA2-specific CD4+/ CD8+ T cell responses. | <ul> <li>CMI response <ul> <li>NTHi-specific and Mcat-specific CMI responses as measured by flow cytometry ICS (frequency of specific CD8+ T-cells expressing at least 2 different markers among CD40L,IL-2, IL-13, IL-17, IFN-γ, TNF-α upon in vitro stimulation) before Dose 1 (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group) in the CMI response sub-cohort.¹</li> </ul> </li> <li>T-helper profile <ul> <li>T-helper profile of the specific T-cell response in T-helper 1, T-helper 2 and T-helper 17 based on the specific expression of respectively IFN- γ, IL-13 and IL-17 before Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group) in the CMI subcohort. Frequencies of specific CD4+/CD8+ T cells per 10<sup>6</sup> cells expressing combinations of</li> </ul> </li> </ul> |

Given the different intervals between vaccines, the label for study visits or contacts varies between treatment groups and as such the Visit/contact label varies. Please refer to the study design diagram (Figure 1).

<sup>&</sup>lt;sup>2</sup> Cut-off for seropositivity will be the lower limit of quantification (LLOQ) of the assay.

<sup>&</sup>lt;sup>3</sup> Refer to Section 5.3.1 of the study protocol for details regarding the CMI sub-cohort.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

### 4. ANALYSIS SETS

### 4.1. Definition

| Analysis Set | Description |
|---|---|
| Enrolled All subjects who signed informed consent | |
| Exposed (ES) All subjects who received at least 1 dose of the study treatment. The in a group is done in function of the administered treatment. | |
| Full analysis (FAS) | All subjects who received at least 1 dose of the study treatment and have post-vaccination immunogenicity data |
| Modified full analysis (mFAS) All subjects who received full study treatment course to which they are randomized and have post-vaccination immunogenicity data | |
| Per protocol (PPS) All subjects who received full study treatment course to which the randomized and have post-vaccination data (mFAS) minus subject protocol deviations that lead to exclusion | |
| Unsolicited safety | All subjects who received at least 1 dose of the study treatment¹ (exposed set) that report unsolicited AEs or that report not having unsolicited AEs |
| Solicited safety | All subjects who received at least 1 dose of the study treatment¹ (exposed set) who have solicited safety data |

<sup>1</sup> Study treatment refers to the NTHi-Mcat vaccine. Please refer to Section 4.1.1 for additional details.

#### 4.1.1. Additional considerations

The Enrolled set includes all subjects who signed informed consent, excluding subjects withdrawn prior to randomization (e.g. screening failures).

For the Unsolicited and Solicited safety sets, 1 dose of the study treatment refers to the administration of at least 1 dose of the NTHi-Mcat vaccine, in line with the study analysis of solicited and unsolicited AEs. In addition, subjects exposed to *Shingrix* only (if any) will be included in an extra group named "Shingrix only" for the safety analyses based on the Exposed Set (ES). Refer to Section 9.1.2 for more details about the algorithm to attribute subjects to groups for the purpose of safety analyses.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Details are provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (study vaccine not administered at all), code 800 (fraudulent data) and code 900 (invalid informed consent) will be used for identifying subjects eliminated from the ES.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

Subjects assigned to code 1030.b (not administering any NTHi-Mcat vaccine), but not to code 1030 will be identified as subjects belonging to the "Shingrix only" group.

## 4.2.2. Elimination from Full analysis set (FAS)

### 4.2.2.1. Excluded subjects

A subject will be excluded from the FAS analysis under the following conditions:

| Code | Condition under which the code is used | Visit (V) (timepoints) where the code is applicable | Applicable for endpoint [HUM=humoral response, CMI=CMI response] |
|---|---|---|---|
| 800 | Fraudulent data | All | HUM, CMI |
| 900 | Invalid informed consent | All | HUM, CMI |
| 1030 | Study vaccine not administered at all | All | HUM, CMI |
| 2100.a | Humoral immune response results not available post-vaccination | V6_1, V6_3, V6_6, V4 | HUM |
| 2100.b | CMI response results not available post-vaccination | V6_1, V6_3, V6_6, V4 | CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

Note: in case a subject is bled but blood sample is not planned per study protocol (code 2130), the unexpected sample is eliminated from the analysis, but subject is retained.

## 4.2.3. Elimination from Modified full analysis set (mFAS)

### 4.2.3.1. Excluded subjects

A subject will be excluded from the mFAS analysis <u>if excluded from the FAS</u> and under the following additional conditions:

| Code | Condition under which the code is used | Visit (V) (timepoints) where the code is applicable | Applicable for endpoint [HUM=humoral response, CMI=CMI response] |
|---|---|---|---|
| 1030.b | Not administering any NTHi-Mcat vaccine | All | HUM, CMI |
| 1070.a | Incomplete treatment course | All | HUM, CMI |
| 1070.a | Other deviations related to wrong treatment administered (including randomization failure) | All | HUM, CMI |
| 2080 | Subjects did not comply with Sh_NTHi-<br>Mcat vaccination schedule | V3_1, V3_3, V3_6 | HUM, CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## 4.2.4. Elimination from Per-protocol analysis set (PPS)

## 4.2.4.1. Excluded subjects

A subject will be excluded from the PPS analysis <u>if excluded from the mFAS</u> and under the following additional conditions:

| Code | Condition under which the code is used | Visit (V)<br>(timepoints)<br>where the code<br>is applicable | Applicable for endpoint<br>[HUM=humoral<br>response, CMI=CMI<br>response] |
|---|---|---|---|
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol | All | HUM, CMI |
| 1070 | Vaccination not according to protocol | All | HUM, CMI |
| 1080 | Vaccine temperature deviation | All | HUM, CMI |
| 1090 | Expired vaccine administered | All | HUM, CMI |
| 2010 | Protocol violation (inclusion/exclusion criteria) | All | HUM, CMI |
| 2040 | Administration of any medication forbidden by the protocol | All | HUM, CMI |
| 2050 | Medical condition forbidden by the protocol | All | HUM, CMI |
| 2080 | Subjects did not comply with vaccination schedule | All | HUM, CMI |
| 2090.a | Subjects did not comply with blood sample schedule (sample for humoral immune response) | All | HUM |
| 2090.b | Subjects did not comply with blood sample schedule (sample for CMI response) | All | CMI |
| 2100.a | Humoral immune response results not available | All | HUM |
| 2100.b | CMI response results not available | All | CMI |
| 2120.a | Obvious incoherence or abnormality or error in data (data on humoral immune response) | All | HUM |
| 2120.b | Obvious incoherence or abnormality or error in data (data on CMI response) | All | CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

## 4.2.5. Elimination from unsolicited and solicited safety set

## 4.2.5.1. Excluded subjects

## 4.2.5.1.1. Unsolicited safety set

Code 1030.b (not administering any NTHi-Mcat vaccine), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1150 (no post-vaccination safety data) will be used to identify subjects eliminated from the unsolicited safety set.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

Code 1150 will be attributed to subjects if <u>all</u> the following conditions are met: subject did not complete the safety assessment following the 7-day follow-up period after NTHi-Mcat vaccinations (i.e. phone contacts), did not return the pDiary, did not return for the scheduled visit 30-days after the NTHi-Mcat vaccinations and did not report any unsolicited AE.

Code 1070.a will be used to identify subjects eliminated from the Unsolicited Safety Set by visit when the NTHi-Mcat vaccination is not administered at that visit.

### 4.2.5.1.2. Solicited safety set

Code 1030.b (not administering any NTHi-Mcat vaccine), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data) will be used to identify subjects eliminated from the solicited safety set.

Code 1070.a will be used to identify subjects eliminated from the Solicited Safety Set by visit when the NTHi-Mcat vaccination is not administered at that visit.

### 5. STATISTICAL ANALYSES

Note that standard data derivation rules and statistical methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and statistical methods will be described in Section 9.

# 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (including age at first study vaccination in years, gender, race, ethnicity and smoking status) will be summarized by study group and overall, using descriptive statistics:

- Frequency tables will be generated for categorical variables such as smoking status.
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age, height and weight.

Withdrawal status will be summarized by group using descriptive statistics:

- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal
- The number of subjects enrolled into the study as well as the number of subjects excluded from the PPS and mFAS will be tabulated.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

### 5.1.2. Additional considerations

Summaries of demographic/baseline characteristics will include: age, country, centre, gender, race, ethnicity, smoking status, pack-years and vital signs (including body mass index [BMI]).

# 5.2. Exposure

## 5.2.1. Analysis of exposure planned in the protocol

None.

#### 5.2.2. Additional considerations

The number and percentage of subjects who received study vaccine doses will be tabulated for each study group (based on the ES).

## 5.3. Immunogenicity

## 5.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PPS. A supplementary analysis may be based on the mFAS.

| Endpoint | Statistical analysis methods |
|---|---|
| Primary | Between group assessment Considering the sampling timepoint at 1 month after Dose 2 of NTHi-Mcat vaccine, the 2-sided 95% CIs for the group GMC ratio (Sh_NTHi-Mcat_1; _3; _6 group over NTHi-Mcat group) of anti-PD, anti-PE, anti-PilA, anti-UspA2 will be computed using an analysis of covariance (ANCOVA) model on the logarithm10 transformation of the concentrations. The ANCOVA model will include study group, smoking status (current or former), age category (50–59, 60–69, 70–80 years of age) and centre as factors and the antibody concentration before Dose 1 as covariate. |
| | Non-inferiority for a specific time-lag will be claimed if the lower limit of the 2-sided 95% CI for the GMC ratio will be above 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2. The sequential procedure for multiple time-lags will be used: starting from the 6-months lag, the 3-months NI will be tested only if the 6-months NI will be demonstrated, while the 1-month NI will be tested only if the 6-months and 3-months NI will be both demonstrated. |
| Secondary - humoral | Within group assessment For each study group, for each sampling timepoint and for each antigen, the following statistics will be computed: Seropositivity rates with exact 95% CI (seropositivity defined using the assay lower limits of quantification [LLOQ]) Adjusted and unadjusted GMCs with 95% CI (adjustment by ANCOVA model, as specified above) The range and distribution of antibody concentrations The distribution of antibody concentrations for each antigen will be displayed using reverse cumulative distribution curves. |

30-JAN-2020 17

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

| Endpoint | Statistical analysis methods |
|---|---|
| Secondary –cell-<br>mediated immune<br>response | CMI response induced by the NTHi-Mcat candidate vaccine will be evaluated, presenting the frequencies of antigen-specific CD4+ T cells per 10 <sup>6</sup> cells. The specific CD4+ T cells being identified as the CD4 + T cells expressing at least 2 different markers among CD40 Ligand (CD40L), IL-2, TNF- α, IFN- γ, IL-13 and IL-17 upon in vitro stimulation. Descriptive statistics (Min, Q1, Median, Mean, Q3 & Max) will be reported for each group at pre-Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh-NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group). |
| Tertiary -cell-<br>mediated immune<br>response | <ul> <li>CMI response induced by the NTHi-Mcat candidate vaccine will be evaluated, presenting the frequencies of antigen-specific CD8+T cells per 10<sup>6</sup> cells. The specific CD8+T cells being identified as the CD8+ T cells expressing at least 2 different markers among CD40L, IL-2, TNF- α, IFN- γ, IL-13 and IL-17 upon in vitro stimulation.</li> <li>CMI response as the frequencies of specific CD4+/CD8+ T cells per 10<sup>6</sup> cells expressing any combination of cytokines/activation markers will be determined. The T-helper profile of the specific T-cell response in T-helper 1, T-helper 2 and T-helper 17 based on the specific expression of respectively IFN-γ, IL-13 and IL-17 will be characterized.</li> <li>Descriptive statistics (Min, Q1, Median, Mean, Q3 &amp; Max) will be reported for each group at pre-Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh-NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group).</li> </ul> |

#### 5.3.2. Additional considerations

The supplementary analysis based on the mFAS will be performed if the percentage of mFAS subjects excluded from the PPS is more than 10%.

#### 5.3.2.1. Analysis of humoral response

## Hypothesis related to the primary objective

The global null hypothesis related to the primary objective of the study is that at least 1 GMC ratio (Sh\_NTHi-Mcat over NTHi-Mcat) among anti-PD, anti-PE, anti-PilA, anti-UspA2 is inferior or equal to 0.667 in all time-lags under investigation at 1 month post-Dose 2 of NTHi-Mcat vaccine. This must be rejected in favour of the alternative hypothesis that all 4 GMCs (anti-PD, anti-PE, anti-PilA, anti-UspA2) are non-inferior in at least one time-lag group. Family-wise type I error is fixed at 2.5% (1-sided).

## Geometric mean concentration and geometric mean concentration ratio

For each antigen and study group, at 1 month after Dose 2 of NTHi-Mcat vaccine, adjusted GMCs and GMCs ratios with corresponding 95% CIs will be obtained exponentiating (base 10) the least square means and the lower and upper limits of the 95% CIs derived from the ANCOVA model. The ANCOVA model will be implemented in SAS, similarly to the following code:

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

```
PROC GLM data=<dataset>;
BY antigen;
class group age smoking_status centre;
MODEL log(concentr) = group age smoking_status centre log(pre_concentr);
LSMEAN group / CL PDIFF ALPHA=0.05;
RUN;
```

Contrasts to be included: Sh\_NTHi-Mcat\_6 vs NTHi-Mcat, Sh\_NTHi-Mcat\_3 vs NTHi-Mcat, Sh\_NTHi-Mcat\_1 vs NTHi-Mcat.

In addition, unadjusted GMCs and GMRs will be presented for each timepoint (pre-Dose 1 and post-Dose 2 of NTHi-Mcat vaccine) with a descriptive purpose.

## Permutation test (sensitivity analysis on primary objectives)

Based on the covariate-adaptive treatment assignment algorithm (see Section 10.3), the following permutation test will be performed as a sensitivity analysis on the primary objectives [Wiens, 2006, Hasegawa, 2009 and Ernst, 2004] in the PPS.

For each antigen, let  $\mathbf{X}=(X_1,\ldots,X_N)$  the logarithmically-transformed antibody concentrations for the NTHi-Mcat group and  $\mathbf{Y}_{1/3/6}=(Y_1,\ldots,Y_N)$  the logarithmically-transformed antibody concentrations for one of the Sh\_NTHi-Mcat groups at 1 month after Dose 2 of NTHi-Mcat vaccine, a non-inferiority permutation test can be obtained from a superiority permutation test on  $\dot{\mathbf{X}}=(X_1,\ldots,X_N)$  against  $\dot{\mathbf{Y}}_{1/3/6}=(Y_1+\delta,\ldots,Y_N+\delta)$  with  $\delta=0.176=-\log_{10}(0.667)$ .

The original treatment assignment algorithm will be used to re-randomize subjects while keeping antibody concentrations, covariates and entry order as observed. The procedure will be as follows:

- 1. Fit the ANCOVA model to obtain the test statistics  $T*_{1/3/6}$  for the superiority of  $\dot{\mathbf{X}}$  against  $\dot{\mathbf{Y}}_{1/3/6}$ .
- 2. Estimate the distribution of the test statistics with R=10000 repetitions of the following 2 steps:
  - a. Re-randomize treatment assignment of all 4 groups (original algorithm).
  - b. Re-fit the ANCOVA model to re-obtain the test statistics  $T_{1/3/6}$ .
- 3. Derive the permutation p-values associated to the observed test statistics (from step 1) based on the empirical distributions in Step 2

$$\mathbf{p}_{1/3/6} = \mathbf{M} + 1/\mathbf{R} + 1$$

Where M is the number of repetitions such that  $T_{1/3/6} \ge T^*_{1/3/6}$ .

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

#### Seropositivity rate and fold increase

For each antigen, timepoint and study group, the seropositivity rate (defined as the proportion of subjects with an antibody concentration greater or equal to the assay cut-off) with exact 95% CIs will be computed using the method referenced in section 10.1.5.1. Assay cut-offs are reported in section 9.1.1. In addition, percentages of subjects with a 2/4/8-fold increase will be presented with associated 95% CI.

#### **Reverse cumulative distribution curves**

Reverse cumulative distribution (RCD) curves for antibody concentrations will be plotted: the x-axis represents the antibody concentrations value (log-10 scale), while the y-axis the percentage of subjects having a log-transformed antibody value greater or equal to the corresponding x-value.

### 5.3.2.2. Analysis of CMI response

The frequency of **antigen-specific** CD4+ or CD8+ T-cells for each individual subject is calculated as the difference between the frequency of CD4+ or CD8+ T-cells producing at least 2 activation markers among CD40 Ligand (CD40L), IL-2, TNF-  $\alpha$ , IFN-  $\gamma$ , IL-13 and IL-17, upon *in vitro* stimulation with the antigen (induction condition) minus the frequency of CD4+ or CD8+ T-cells producing at least 2 activation markers upon in vitro stimulation in medium only (background condition). For descriptive statistics purposes, differences less or equal to zero (0) are imputed to 1.

# 5.4. Analysis of safety and reactogenicity

# 5.4.1. Analysis of safety and reactogenicity planned in the protocol

All safety analyses will be performed on the solicited safety set, unsolicited safety set and exposed set.

| Endpoint | Statistical analysis methods |
|---|---|
| Secondary | Within group assessment The percentage of subjects with at least 1 local adverse event (AE) (solicited and unsolicited), with at least 1 general AE (solicited and unsolicited) and with any AE during the 7-days solicited follow-up period and the 30-days follow-up period will be tabulated by group with exact 95% CI after each NTHi-Mcat vaccine dose and overall. The percentage of NTHi-Mcat doses followed by at least 1 local AE (solicited and unsolicited), by at least 1 general AE (solicited and unsolicited) and by any AE will be tabulated by group with exact 95% CI. The same calculations will be performed for AEs rated as Grade 3, for AEs causally related to vaccination and Grade 3 AEs causally related to vaccination. |
| | The percentage of subjects reporting each individual solicited local and general AE during the 7-days solicited follow-up period after each dose of NTHi-Mcat vaccine will be tabulated by group with exact 95% CI. The percentage of NTHi-Mcat doses followed by each individual solicited local and general AE will be tabulated by group with exact 95% CI. Fever will be reported per 0.5°C cumulative increments. For all solicited symptoms, the same tabulation will be performed for Grade 3 AEs. The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) |

30-JAN-2020 20

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

| Endpoint | Statistical analysis methods |
|---|---|
| | Dictionary for Adverse Event Terminology. The percentage of subjects with at least 1 report of unsolicited adverse event classified by the MedDRA and reported up to 30 days after NTHi-Mcat vaccinations will be tabulated by group with exact 95% CI. The same tabulation will be performed for Grade 3 unsolicited adverse events, for unsolicited adverse events with a causal relationship to vaccination and for Grade 3 AEs causally related to vaccination. |
| | The number of subjects who experienced any serious adverse event (SAE) or any potential immune-mediated disease (pIMD) from Day 1 to Day 331 and from Day 331 to Day 661 will be reported. |
| | The number of subjects who experienced any AE leading to study withdrawal, from first vaccination up to study conclusion, or any SAE related to study participation or concurrent GSK medication/vaccination, during the entire study period, will be reported. |
| | A summary of subjects reporting concomitant medication/product will be provided. |

#### 5.4.2. Additional considerations

## 5.4.2.1. Analysis of solicited AEs

The analysis of solicited AEs will be performed on the Solicited safety set.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals as follows:

Grade 0: <20 mm diameter

Grade 1: ≥20 mm to ≤50 mm diameter

Grade 2: >50 mm to ≤100 mm diameter

Grade 3: >100 mm diameter

Temperature (i.e. fever) will be scored at GSK Biologicals as follows:

Grade 0: <37.5°C

Grade 1: 37.5°C to 37.9°C

Grade 2: 38.0°C to 38.9°C

Grade  $3: \ge 39.0$ °C

Fever, defined as a body temperature of  $\geq$ 37.5°C irrespective of route of measurement, will be integrated to the summaries as a general AE.

In addition, body temperature will be broken down into 0.5°C increments:

- <36.0
- -36.0 36.4
- -36.5 36.9
- -37.0-37.4
- -37.5 37.9
- -38.0 38.4
- -38.5 38.9
- -39.0 39.4
- -39.5 39.9
- >40.0

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

Compliance of subjects in completing solicited AEs information will be reported as the percentage of subjects completing at least 80% of the diary entries related to local and general solicited AEs.

#### 5.4.2.2. Analysis of unsolicited AEs

The analysis of unsolicited AEs will be performed on the Unsolicited safety set.

Analysis of unsolicited AEs will be also stratified on AEs with a causal relationship to NTHi-Mcat vaccination.

## 5.4.2.3. Combined analysis of solicited and unsolicited AEs

The combined analysis of solicited and unsolicited AEs will be performed on the Unsolicited safety set.

Solicited AEs will be coded by MedDRA as per the following codes:

| Solicited symptom | Preferred Term code | Corresponding Preferred Term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Redness | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Gastrointestinal symptoms | 10017944 | Gastrointestinal disorder |
| Myalgia | 10028411 | Myalgia |
| Chills | 10008531 | Chills |
| Fever | 10037660 | Pyrexia |

Combined analysis of solicited and unsolicited AEs will be also stratified on AEs with a causal relationship to NTHi-Mcat vaccination (all solicited AEs are considered causally related).

## 5.4.2.4. Analysis of SAEs and pIMDs

The analysis of SAEs and pIMDs will be performed on the Exposed Set (ES).

Analysis of SAEs will include:

- All SAEs from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
- Fatal SAEs from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
- Related SAEs:
  - To any study vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.

22

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

- To the NTHi-Mcat vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661, from the day of the first NTHi-Mcat vaccination up to 1 month following the second dose, from the day of the first NTHi-Mcat vaccination up to 6 months following the second dose and from the day of the first NTHi-Mcat vaccination up to 12 months following the second dose (all groups except "Shingrix only").
- To Shingrix vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661 (all groups except NTHi-Mcat).

Analysis of pIMDs will include all occurrences from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.

## 5.4.2.5. Other safety analyses

Medications will be coded using GSKDRUG dictionary.

All collected concomitant medications and vaccinations will be listed. In addition, prior and concomitant vaccinations will be summarized. In case of pregnancies during the study, follow-up data and pregnancy outcomes will be described in detail.

### 6. ANALYSIS INTERPRETATION

Except for analysis on primary objectives, with predefined success criteria and an appropriate type I error control, comparative analyses are descriptive with the aim to characterize the difference between groups.

With respect to confirmatory analyses on primary objectives the interpretation will be done in a hierarchical manner.

Each objective can only be reached if all the associated criteria are met and all previous objectives have been reached (see Figure 2): starting from the 6-months lag, the 3-months NI can be achieved only if the 6-months NI is demonstrated, while the 1-month NI can be achieved only if the 6-months and 3-months NI are both demonstrated.

This sequential procedure enables to control the overall type I error below 2.5% (one-sided) [Dmitrienko, 2009].

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

Figure 2 Sequence for evaluating the primary objective in order to control the overall type I error below 2.5% (one-sided)



## 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

The integrated clinical study report (CSR) will contain at least the final analyses of all primary and secondary endpoints. If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These analyses will be documented in annex(es) to the study report.

The analyses will be performed stepwise:

- A final analysis of immunogenicity, safety and reactogenicity for all subjects up to and including Day 331 ('Epoch 001') will be performed in a first step.
  - A complete study report containing all data of 'Epoch 001' will be written and made available to the investigators at this stage.
- Analysis conducted on the data collected for all subjects from Day 331 up to and including Day 661 ('Epoch 002') will be performed in a second step.

An integrated CSR containing all data from Epoch 001 and Epoch 002 will be written and made available to the investigators.

| Description | Disclosure Purpose |
|---|---|
| | (CTRS=public posting, SR=study report, internal) |
| Final Analysis Epoch 001 | Web disclosure (CTRS), Study report (SR) |
| Analysis of Follow-up Epoch | Web disclosure (CTRS), Study report (SR) |

# 7.2. Statistical considerations for interim analyses

No interim analysis is planned for this study. Data up to and including Day 331 are considered 'final' and completed data, while the remaining safety data are considered long-term safety follow-up.

24

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## 8. CHANGES FROM PLANNED ANALYSES

Not applicable

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in Section 10.1

### 9.1. Data derivation

## 9.1.1. Assay cut-offs for serology results

| Component | Method | Unit <sup>1</sup> | Assay cut-off <sup>1</sup> |
|---|---|---|---|
| anti-PD antibody | ELISA | EU/mL | 153 |
| anti-PE antibody | ELISA | EU/mL | 25 |
| anti-PilA antibody | ELISA | EU/mL | 16 |
| anti-UspA2 IgG antibody | ELISA | EU/mL | 38 |

ELISA = Enzyme Linked Immunosorbent Assay; EU/ml = ELISA unit per millilitre; Ig = immunoglobulin; PD = protein D; from NTHi; PE = protein E from NTHi; PilA = type IV pili subunit from NTHi; UspA2 = ubiquitous surface protein A2 from Mcat

# 9.1.2. Attributing subjects to time-lag groups

For the purpose of safety analyses, the following rule will be used to attribute exposed subjects to a specific group.

- If a subject receives no *Shingrix* vaccination → NTHi-Mcat group
- If a subject receives at least 1 Shingrix vaccination, but no NTHi-Mcat vaccination
   → "Shingrix only" group
- If a subject receives at least 1 *Shingrix* vaccination and at least 1 NTHi-Mcat vaccination, the difference, in days, between the latest Shingrix vaccination and the earliest NTHi-Mcat vaccination will be computed and converted in months (diff):
  - $diff ≤ 2 \rightarrow Sh_NTHi-Mcat_1 group$
  - 2 < diff ≤ 4.5  $\rightarrow$  Sh\_NTHi-Mcat\_3 group
  - diff > 4.5  $\rightarrow$  Sh NTHi-Mcat 6 group

#### 9.2. Statistical Method

Not applicable

<sup>1</sup> Assay cut-off and unit might be subject to change during the course of the study (e.g. in case of assay reoptimization, qualification, (re)validation or standardization). In this case, this will be documented in the clinical study report.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in Section 9 (additional study-specific rules).

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the eCRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30th.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

#### 10.1.2.3. Daily recording of solicited symptoms

### 10.1.2.3.1. Studies with paper diaries

Denominators for the summary of local (or general) solicited symptoms will be calculated using the number of subjects who respond "Yes" or "No" to the question concerning the occurrence of local (or general) symptoms.

When a specific symptom is marked as having not occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=N for the specified post-vaccination period for the symptom in question), all daily measurements will be imputed as Grade 0.

When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

When the occurrence of a specific symptom is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-vaccination period for the symptom in question) but the group of symptoms (local or general) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

The following table shows how subjects contribute to each category for a specific solicited symptom over the Day X to Day Y post-vaccination period:

| Solicited symptom category | Subjects included in the calculation of the numerator |
|---|---|
| Any | All subjects with at least one occurrence of the symptom at Grade 1, Grade 2, or Grade 3 between Day X and Day Y or with the symptom marked as present and at least one missing daily recording between Day X and Day Y |
| At least Grade 1 | All subjects with at least one occurrence of the symptom at Grade 1, Grade 2, or Grade 3 between Day X and Day Y |
| At least Grade 2 | All subjects with at least one occurrence of the symptom at Grade 2 or Grade 3 between Day X and Day Y |
| At least Grade 3 | All subjects with at least one occurrence of the symptom at Grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### 10.1.3. Data derivation

### 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years

DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

## 10.1.3.2. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (weight in kilograms) / (height in meters) $^2$ 

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

#### 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

### 10.1.3.4. Geometric mean concentrations (GMCs)

GMC calculations are performed by taking the inverse logarithm of the mean of the log-10 concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

#### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus 1 day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the consecutive days with the symptom reported at Grade 1 or higher. The duration of solicited events at a specific grade (e.g. Grade 3) will be calculated as the sum of the consecutive days with the symptom reported at that grade. The same rule applies for solicited events ongoing at the end of the solicited follow-up period considering the maximum intensity reported.

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event eCRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

### 10.1.3.8. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarised, each event recorded as having occurred during a specific period will be counted as the number of occurrences the event is consecutively reported (at Grade 1 or higher). When the occurrences of solicited adverse events at a specific grade are summarised, each event recorded as having occurred at that grade during a specific period will be counted as the number of occurrences the event is consecutively reported at that grade.

## 10.1.4. Display of decimals

## 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

30

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

#### 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with 1 more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with 1 decimal will be displayed with 2 decimals.

#### 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, BMI, pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height variables will be displayed with no decimals.

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values below 10kg where 1 decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with 1 decimal.

## 10.1.4.4. Serological summary statistics

The number of decimals used when displaying GMCs and their confidence limits is shown in the following table:

| GMC value | Number of decimals to display |
|----------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the 1 with the higher number of decimals). For example, if GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

31

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

## 10.1.5. Statistical methodology

#### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Mietinnen and Nurminen [Miettinen, 1985].

#### 10.1.5.3. Adjusted GMC ratios

When between-group GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure.

## 10.2. TFL ToC

The list of tables, figures and listings (TFL ToC) planned for this study can be found in eTMF folder section 11.1.1

## 10.3. Randomization method and minimization algorithm

The minimization algorithm used at the GSK internet randomization system (i.e. SBIR) for study NTHI MCAT-009 is based on the following reference: "White SJ, Freedman LS. Allocation of patients to treatment groups in a controlled clinical study. Br J Cancer 1978; 37: 849-857" [White, 1978] and it is described below:

#### **Notations**

- K=3 input values [Centre, Smoking status and Age category] to be used for minimization, each with a weight  $w_k=1$  (k=1,...,K) &  $l_k$  variants.
- I=4 treatment groups [NTHi-Mcat, Sh\_NTHi-Mcat\_6, Sh\_NTHi-Mcat\_3, Sh\_NTHi-Mcat\_1] with randomization ratio a<sub>1</sub>,...,a<sub>I</sub> [1:1:1:1]

32

#### Algorithm

For a new subject with input value variants  $s_1...s_K$ 

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## Step 1: Minimization computation

Step 1.1: Initialize Problem flag to 0

For each input value variant  $s_k$ , compute the number of subjects already enrolled in each treatment group.

Let  $b_{ik}$  the number for treatment i & input value variant  $s_k$ :  $b_{ik}$  is the total number of subjects already randomized in treatment i and with variant  $s_k$ .

Step 1.2: For each treatment i: compute  $A_i = 1/a_i * sum_k(w_k * b_{ik})$ 

Step 2: determine whether the algorithm is random or deterministic:

Generate R, a random number within [0-1], uniform distribution

Step 3: check determinism

If R < 0.9, go to step 4 (determinism) else go to step 5 (random)

Step 4: determinism

4.1: Identify all treatments with the lowest value A<sub>i</sub>

4.2: Select randomly one of the treatments identified in step 4.1, let it be T.

Go to step 6, if no more treatment then randomization failed

Step 5: randomization

Select randomly one of the treatments, let it be T.

Go to step 6, if no more treatment then randomization failed.

Step 6: treatment allocation

Assign one of the treatment nr. related to treatment T in the subject's center.

If no treatment nr. related to treatment T is available in the subject's center, then go & repeat step 4 (determinism) or 5 (random) while dropping treatment T (set problem flag=1).

209538 (NTHI MCAT-009) Statistical Analysis Plan Amendment 1

## 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934; 26:404-13.

Dmitrienko, A., Tamhane, A. C., & Bretz, F. (2009). Multiple testing problems in pharmaceutical statistics. CRC press.

Ernst MD, Permutation Methods: A Basis for Exact Inference. *Statistical Science*, 2004; 19: 676-685.

Hasegawa T, Tango T. Permutation test Following Covariate-Adaptive Randomization in Randomized Controlled Trials. *Journal of Biopharmaceutical Statistics*, 2009; 19: 106-119.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. *Statistics in Medicine*, 1985;4:213-226.

White SJ, Freedman LS. Allocation of patients to treatment groups in a controlled clinical study. *Br J Cancer*, 1978;37: 849-857

Wiens BL, Randomization as basis for inference in noninferiority trials. *Pharmaceutical Statistics*, 2006; 5: 265-271

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

| | Statistical Analysis Plan Fina |
|---|---|
| GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | Immunogenicity and safety study of GSK's investigational vaccine (GSK3277511A) when administered in healthy smokers and ex-smokers following receipt of <i>Shingrix</i> vaccine. |
| eTrack study number and<br>Abbreviated Title | 209538 (NTHI MCAT-009) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 01 April 2019 |
| Co-ordinating author: | (Statistician) |
| Reviewed by: | <ul> <li>PPD (Clinical &amp; Epidemiology Project Lead)</li> <li>PPD (Clinical Research &amp; Development Lead)</li> </ul> |
| | <ul> <li>PPD (Lead Statistician)</li> <li>PPD (Lead Statistical Analyst)</li> <li>PPD (Statistical Analyst)</li> <li>PPD (Scientific writer)</li> <li>PPD (Stat Peer Reviewer)</li> </ul> |
| | <ul> <li>PPD (Regulatory Affairs)</li> <li>PPD (SERM scientist)</li> <li>PPD (Public disclosure representative)</li> </ul> |
| Approved by: | <ul> <li>PPD (Clinical &amp; Epidemiology Project Lead)</li> <li>PPD (Clinical Research &amp; Development Lead)</li> <li>PPD (Lead Statistician)</li> <li>PPD (Statistician)</li> <li>PPD (Scientific writer)</li> <li>PPD (Lead Statistical Analyst)</li> </ul> |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 12th November 2018)
209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | | | | | PAGE |
|---|---|---|---|---|---|---|---|
| LIS | T OF A | ABBREVIA | TIONS | | | | 4 |
| 1. | DOC | JMENT HI | STORY | | | | 7 |
| 2. | STUE | Y DESIGN | ١ | | | | 7 |
| 3. | OBJE | CTIVES A | ND ENDP | OINTS | | | 9 |
| 4. | ANAL | YSIS SET | S | | | | 11 |
| | 4.1. | Definition 4.1.1. | | | | | |
| | 4.2. | | | | | | |
| | | 4.2.1. | Eliminatio | n from Expos | sed Set (ES) | | 11 |
| | | 4.2.2. | Eliminatio | n from Full a | nalysis set (FAS | ) | 12 |
| | | | 4.2.2.1. | Excluded s | ubjects | | 12 |
| | | 4.2.3. | | | | set (mFAS) | |
| | | | 4.2.3.1. | Excluded s | ubjects | | 12 |
| | | 4.2.4. | | n from Per-p | rotocol analysis | set (PPS) | 13 |
| | | | 4.2.4.1. | | | | |
| | | 4.2.5. | | | | ed safety set | |
| | | | 4.2.5.1. | | | | |
| | | | | | | ety set | |
| | | | | 4.2.5.1.2. | Solicited safety | v set | 14 |
| 5. | STAT | ISTICAL A | NALYSES | | | | 14 |
| ٠. | 5.1. Demography | | | | | | |
| | | 5.1.1. | Analysis c | of demograph | ics/baseline cha | aracteristics plann | ed |
| | | 5.1.2. | | | | | |
| | 5.2. | | | | | | |
| | 0.2. | 5.2.1. | | | | otocol | |
| | | 5.2.2. | | | | | |
| | 5.3. | | | | | | |
| | 0.0. | 5.3.1. | | | | the protocol | |
| | | 5.3.2. | Additional | consideration | ns | | 16 |
| | | | 5.3.2.1. | | | se | |
| | | | 5.3.2.2. | | | | |
| | 5.4. | Analysis | | | | | |
| | | 5.4.1. | • | • | reactogenicity p | | |
| | | | | | | | 18 |
| | | 5.4.2. | | | | | |
| | | | 5.4.2.1. | Analysis of | solicited AEs | | 19 |
| | | | 5.4.2.2. | | | | |
| | | | 5.4.2.3. | Combined a | analysis of solicit | ted and unsolicite | d |
| | | | 5.4.2.4. | | | S | |
| | | | 5.4.2.5. | | | | |
| | | | J. 1.2.J. | Julior Juliot | , analyses | | |
| 6 | ANAI | YSIS INTE | RPRETAT | ΓΙΟΝ | | | 21 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Final CONDUCT OF ANALYSES......22 Sequence of analyses.....22 7.2. CHANGES FROM PLANNED ANALYSES......22 NON-STANDARD DATA DERIVATION RULES AND STATISTICAL 9. 9.1. Data derivation ......23 Attributing subjects to time-lag groups .......23 9.1.2. 9.2. Statistical Method 23 10. ANNEXES \_\_\_\_\_\_\_24 10.1. Business rules for standard data derivations and statistical methods.......24 10.1.1. Attributing events to vaccine doses......24 10.1.2. Handling of missing data.....24 Dates.....24 Laboratory data ......25 10.1.2.2. 10.1.2.3. Daily recording of solicited symptoms......25 10.1.2.4. 10.1.3. 10.1.3.2. Body mass index (BMI) ......26 Numerical serology results ......27 10.1.3.3. 10.1.3.4. Geometric mean concentrations (GMCs)......27 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events ......28 Counting rules for occurrences of solicited 10.1.3.8. adverse events......28 10.1.4. 10.1.4.2. Differences in percentages .......29 Demographic/baseline characteristics statistics......29 10.1.4.3. Statistical methodology......30 10.1.5. 10.1.5.1. Exact confidence intervals around proportions .........30 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions ......30 10.2. 10.3. 

# 209538l Statistical Analysis Plan $\,$ 01 Apr2019l TMF-855396 l2.0

# CONFIDENTIAL

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# **LIST OF TABLES**

| | | PAGE |
|---------|----------------------------------------------------------|------|
| Table 1 | Study groups, treatment and epochs foreseen in the study | 8 |

# 209538l Statistical Analysis Plan $\,$ 01 Apr2019l TMF-855396 l2.0

# CONFIDENTIAL

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design overview | 7 |
| Figure 2 | Sequence for evaluating the primary objective in order to control the overall type I error below 2.5% (one-sided) | 21 |

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# **LIST OF ABBREVIATIONS**

AE Adverse event

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

CI Confidence Interval

CMI Cell-Mediated Immune

eCRF Electronic Case Report Form

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

EU/mL ELISA unit per milliliter

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set

eTMF Electronic Trial Master File

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMR Geometric mean ratio

GSK GlaxoSmithKline

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

NA Not Applicable
NI Non-Inferiority

PD Protocol Deviation

PPS Per-Protocol Set

RCD Reverse cumulative distribution

SAE Serious adverse event

SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SDTM Study Data Tabulation Model

SR Study Report

TFL Tables Figures and Listings

ToC Table of Content

UL Upper Limit of the confidence interval

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|-------------------------|
| 01 APR 2019 | Final version | Protocol Administrative |
| | | Change 1: 14 DEC |
| | | 2018 |

## 2. STUDY DESIGN

Figure 1 Study design overview



BS C = blood sample for cell-mediated immune response; BS H = blood sample for humoral immune responses/assay development from all subjects; C= Call; D = Day; mth(s) = month(s); NA = not applicable; NM = NTHi-Mcat vaccination; RAND = randomization; S = Safety; Sh = Shingrix vaccination; V = Visit

## Notes:

- <sup>1</sup> Groups: Sh NTHi-Mcat 1 (NTHi-Mcat vaccine administered 1 month after *Shingrix* vaccine)
- <sup>2</sup> Groups: Sh\_NTHi-Mcat\_3 (NTHi-Mcat vaccine administered 3 months after *Shingrix* vaccine)
- 3. Groups: Sh\_NTHi-Mcat\_6 (NTHi-Mcat vaccine administered 6 months after Shingrix vaccine)

<sup>&</sup>lt;sup>4.</sup> Patients randomized to the NTHi-Mcat control group will receive the first NTHi-Mcat vaccination at Visit 1 (Day 1) and the second NTHi-Mcat vaccination at Visit 3 (Day 61)

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

- 5. Blood sample for cell-mediated immune response will be taken from approximately 60 subjects (~15 subjects in each group. Refer to Section 5.3.1 of the study protocol for details of the CMI sub-cohort
- 6. Solicited local and general adverse events reported during a 7-day follow-up period after Dose 1 and after Dose 2 of NTHi-Mcat vaccine, and unsolicited adverse events reported during a 30-day follow-up period after Dose 1 and after Dose 2 of NTHi-Mcat vaccine will be collected
- 7. Safety follow-up
- **Primary completion date (PCD):** PCD will be 1 month post-Dose 2 of the NTHi-Mcat investigational vaccine (Day 331, based on Sh\_NTHi-Mcat\_6 treatment group).
- End of Study (EoS): Last subject last visit (Day 661).
- **Study groups:** Approximately 540 eligible subjects who will be randomly assigned to 4 study groups in a (1: 1: 1) ratio (Table 1). Please refer to Section 10.1 of the protocol for details related to the determination of sample size.

Table 1 Study groups, treatment and epochs foreseen in the study

| Study Groups | Number Age | | Treatment name | Epochs<br>(Blinding) | |
|---|---|---|---|---|---|
| Study Groups | subjects | (Min-Max) | Treatment name | Epoch 001<br>(open-label) | Epoch 002<br>(open-label) |
| Sh_NTHi-Mcat_1 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| Sh_NTHi-Mcat_3 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| Sh_NTHi-Mcat_6 | 135 | 50 – 80 years | Shingrix / NTHi-Mcat | • | • |
| NTHi-Mcat | 135 | 50 – 80 years | NTHi-Mcat | • | • |

Sh = Shingrix

- **Treatment allocation:** Subjects will be allocated to a study group using an automated, electronic System Built for Internet Randomization (SBIR). The randomization algorithm will use a minimization procedure accounting for age category (50–59, 60–69, 70–80 years of age), smoking status (current or former smoker), and centre. Minimization factors will have equal weight in the minimization algorithm.
- **Blinding:** open-label.
- **Data collection:** Electronic Case Report Form (eCRF). Telephone contact. Solicited and unsolicited symptoms will be collected using a subject Diary (paper diary [pDiary]).
- Safety monitoring: Subjects will be observed for at least 60 minutes after each NTHi-Mcat vaccination for any immediate reactions. Solicited local and general AEs occurring during a 7-day follow-up period after each NTHi-Mcat vaccination (i.e. the day of vaccination and the 6 subsequent days) and unsolicited AEs occurring during a 30-day follow-up period after each NTHi-Mcat vaccination (i.e. the day of vaccination and the 29 subsequent days), will be reported via diary cards. In addition, subjects will be asked at Phone contacts if there were any safety concerns in the 7-day follow-up period after each NTHi-Mcat vaccination; this information will be recorded via the appropriate section of the eCRF. Finally, safety assessments will be performed during each clinic visit and safety follow-up calls to collect

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

information on AEs leading to withdrawal, serious adverse events (SAEs), SAEs related to study participation or to a concurrent GSK medication/vaccine, pregnancies, potential immune-mediated diseases (pIMDs), throughout the whole study period.

# 3. OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| P | rimary |
| <ul> <li>Confirmatory</li> <li>To demonstrate the non-inferiority (NI) of the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine versus the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine alone.</li> <li>Criterion:</li> <li>Lower limit (LL) of the 2-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio (Sh_NTHi-Mcat/NTHi-Mcat) is above a limit of 0.667 for all anti-PD, anti-PE, anti-PilA, anti-UspA2.</li> </ul> | <ul> <li>Humoral immune response</li> <li>Anti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations 1 month after Dose 2 of NTHi-Mcat vaccine in the Sh_NTHi-Mcat groups (Day 181; Day 241; Day 331) compared to antibody concentrations 1 month after Dose 2 in the NTHi-Mcat group (Day 91).<sup>1</sup></li> </ul> |
| | condary |
| Descriptive To evaluate the safety and reactogenicity profile of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 or 3 or 6 months after Shingrix vaccine or when administered alone. | <ul> <li>Solicited local and general adverse events (AEs) <ul> <li>Occurrence of each solicited local and general adverse event (AE), reported during a 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after Dose 1 and after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine, in all subjects in all groups.</li> </ul> </li> <li>Unsolicited AEs <ul> <li>Occurrence of any unsolicited AEs, reported during a 30-day follow- up period (i.e. day of vaccination and 29 subsequent days) after Dose 1 and after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine, in all subjects in all groups.</li> <li>Serious AEs <ul> <li>Occurrence of any SAE reported from first vaccination (Day 1) to Day 331 in all subjects in all groups.</li> <li>Occurrence of any SAE, reported from Day 331 to Day 661 in all subjects in all groups.</li> <li>Potential immune-mediate diseases (pIMD)</li></ul></li></ul></li></ul> |

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

| Endpoints ral response nti-PD, anti-PE, anti-PilA and anti-UspA2 antibody oncentrations and seropositivity in all subjects efore Dose 1 (Day 91; Day 151; Day 241 in the h_NTHi-Mcat groups and Day 1 in the NTHi-Mcat roup), and 1 month after Dose 2 of NTHi-Mcat accine (Day 181; Day 241; Day 331 in the h_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group). Pesponse ITHi-specific and Mcat-specific CMI responses as neasured by flow cytometry ICS (frequency of pecific CD4+ T-cells expressing at least 2 different narkers among CD40 ligand (CD40L), interleukin L)-2, IL-13, IL-17, interferon gamma (IFN-γ), amour necrosis factor alpha (TNF-α) upon in vitro timulation) before Dose 1 (Day 91; Day 151; Day 41 in the Sh_NTHi-Mcat groups and Day 1 in the ITHi-Mcat group), and 1 month after Dose 2 of ITHi-Mcat vaccine (Day 181; Day 241; Day 331 in |
|---|
| nti-PD, anti-PE, anti-PilA and anti-UspA2 antibody concentrations and seropositivity in all subjects efore Dose 1 (Day 91; Day 151; Day 241 in the h_NTHi-Mcat groups and Day 1 in the NTHi-Mcat roup), and 1 month after Dose 2 of NTHi-Mcat accine (Day 181; Day 241; Day 331 in the h_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group). 1,2 esponse ITHi-specific and Mcat-specific CMI responses as neasured by flow cytometry ICS (frequency of pecific CD4+ T-cells expressing at least 2 different narkers among CD40 ligand (CD40L), interleukin L)-2, IL-13, IL-17, interferon gamma (IFN-γ), umour necrosis factor alpha (TNF-α) upon in vitro timulation) before Dose 1 (Day 91; Day 151; Day 41 in the Sh_NTHi-Mcat groups and Day 1 in the ITHi-Mcat group), and 1 month after Dose 2 of ITHi-Mcat vaccine (Day 181; Day 241; Day 331 in |
| THi-specific and Mcat-specific CMI responses as neasured by flow cytometry ICS (frequency of pecific CD4+ T-cells expressing at least 2 different narkers among CD40 ligand (CD40L), interleukin L)-2, IL-13, IL-17, interferon gamma (IFN-γ), amour necrosis factor alpha (TNF-α) upon in vitro timulation) before Dose 1 (Day 91; Day 151; Day 41 in the Sh_NTHi-Mcat groups and Day 1 in the ITHi-Mcat group), and 1 month after Dose 2 of THi-Mcat vaccine (Day 181; Day 241; Day 331 in |
| ne Sh_NTHi-Mcat groups and Day 91 in the NTHi-<br>lcat group) in the CMI response sub-cohort.1 |
| isat greap) in the enim response our constitu |
| esponse ITHi-specific and Mcat-specific CMI responses as neasured by flow cytometry ICS (frequency of pecific CD8+ T-cells expressing at least 2 different narkers among CD40L,IL-2, IL-13, IL-17, IFN-γ, NF-α upon in vitro stimulation) before Dose 1 Day 91; Day 151; Day 241 in the Sh_NTHi-Mcat roups and Day 1 in the NTHi-Mcat group), and 1 nonth after Dose 2 of NTHi-Mcat vaccine (Day 81; Day 241; Day 331 in the Sh_NTHi-Mcat roups and Day 91 in the NTHi-Mcat group) in the IMI response sub-cohort. The er profile of the specific T-cell response in T-elper 1, T-helper 2 and T-helper 17 based on the pecific expression of respectively IFN-γ, IL-13 and IL-17 before Dose 1 of the NTHi-Mcat pose 2 of ITHi-Mcat group, and 1 month after Dose 2 of ITHi-Mcat investigational vaccine (Day 91; Day 181; Day 441; Day 331 in the Sh_NTHi-Mcat groups and Day 1 in the ITHi-Mcat investigational vaccine (Day 181; Day 441; Day 331 in the Sh_NTHi-Mcat groups and Day 1 in the NTHi-Mcat group) in the CMI sub- |

<sup>&</sup>lt;sup>1</sup> Given the different intervals between vaccines, the label for study visits or contacts varies between treatment groups and as such the Visit/contact label varies. Please refer to the study design diagram (Figure 1). 
<sup>2</sup> Cut-off for seropositivity will be the lower limit of quantification (LLOQ) of the assay.

<sup>&</sup>lt;sup>3</sup> Refer to Section 5.3.1 of the study protocol for details regarding the CMI sub-cohort.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

## 4. ANALYSIS SETS

#### 4.1. Definition

| Analysis Set | Description |
|---|---|
| Enrolled | All subjects who signed informed consent |
| Exposed (ES) | All subjects who received at least 1 dose of the study treatment. The allocation in a group is done in function of the administered treatment. |
| Full analysis (FAS) | All subjects who received at least 1 dose of the study treatment and have post-vaccination immunogenicity data |
| Modified full analysis (mFAS) | All subjects who received full study treatment course to which they are randomized and have post-vaccination immunogenicity data |
| Per protocol (PPS) | All subjects who received full study treatment course to which they are randomized and have post-vaccination data (mFAS) minus subjects with protocol deviations that lead to exclusion |
| Unsolicited safety | All subjects who received at least 1 dose of the study treatment¹ (exposed set) that report unsolicited AEs or that report not having unsolicited AEs |
| Solicited safety | All subjects who received at least 1 dose of the study treatment¹ (exposed set) who have solicited safety data |

<sup>&</sup>lt;sup>1</sup> Study treatment refers to the NTHi-Mcat vaccine. Please refer to Section 4.1.1 for additional details.

#### 4.1.1. Additional considerations

For the Unsolicited and Solicited safety sets, 1 dose of the study treatment refers to the administration of at least 1 dose of the NTHi-Mcat vaccine, in line with the study analysis of solicited and unsolicited AEs. In addition, subjects exposed to *Shingrix* only (if any) will be included in an extra group named "Shingrix only" for the safety analyses based on the Exposed Set (ES). Refer to Section 9.1.2 for more details about the algorithm to attribute subjects to groups for the purpose of safety analyses.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Details are provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (study vaccine not administered at all), code 800 (fraudulent data) and code 900 (invalid informed consent) will be used for identifying subjects eliminated from the ES.

Subjects assigned to code 1030.b (not administering any NTHi-Mcat vaccine), but not to code 1030 will be identified as subjects belonging to the "Shingrix only" group.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# 4.2.2. Elimination from Full analysis set (FAS)

## 4.2.2.1. Excluded subjects

A subject will be excluded from the FAS analysis under the following conditions:

| Code | Condition under which the code is used | Visit (V) (timepoints) where the code is applicable | Applicable for endpoint [HUM=humoral response, CMI=CMI response] |
|---|---|---|---|
| 800 | Fraudulent data | All | HUM, CMI |
| 900 | Invalid informed consent | All | HUM, CMI |
| 1030 | Study vaccine not administered at all | All | HUM, CMI |
| 2100.a | Humoral immune response results not available post-vaccination | V6_1, V6_3, V6_6, V4 | HUM |
| 2100.b | CMI response results not available post-<br>vaccination | V6_1, V6_3, V6_6, V4 | СМІ |
| 2130 | Subject bled but blood sample not planned per study protocol | Elimination is specific<br>to the samples not<br>planned per protocol<br>(subject is retained) | HUM, CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

## 4.2.3. Elimination from Modified full analysis set (mFAS)

## 4.2.3.1. Excluded subjects

A subject will be excluded from the mFAS analysis <u>if excluded from the FAS</u> and under the following additional conditions:

| Code | Condition under which the code is used | Visit (V) (timepoints) where the code is applicable | Applicable for endpoint [HUM=humoral response, CMI=CMI response] |
|---|---|---|---|
| 1070.a | Incomplete treatment course | All | HUM, CMI |
| 1070 | Other deviations related to wrong treatment administered (including randomization failure) | All | HUM, CMI |
| 2080 | Subjects did not comply with Sh_NTHi-<br>Mcat vaccination schedule | V3_1, V3_3, V3_6 | HUM, CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

## 4.2.4. Elimination from Per-protocol analysis set (PPS)

### 4.2.4.1. Excluded subjects

A subject will be excluded from the PPS analysis <u>if excluded from the mFAS</u> and under the following additional conditions:

| Code | Condition under which the code is used | Visit (V)<br>(timepoints)<br>where the code<br>is applicable | Applicable for endpoint [HUM=humoral response, CMI=CMI response] |
|---|---|---|---|
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol | All | HUM, CMI |
| 1070 | Vaccination not according to protocol | All | HUM, CMI |
| 1080 | Vaccine temperature deviation | All | HUM, CMI |
| 1090 | Expired vaccine administered | All | HUM, CMI |
| 2010 | Protocol violation (inclusion/exclusion criteria) | All | HUM, CMI |
| 2040 | Administration of any medication forbidden by the protocol | All | HUM, CMI |
| 2050 | Medical condition forbidden by the protocol | All | HUM, CMI |
| 2080 | Subjects did not comply with vaccination schedule | All | HUM, CMI |
| 2090.a | Subjects did not comply with blood sample schedule (sample for humoral immune response) | All | HUM |
| 2090.b | Subjects did not comply with blood sample schedule (sample for CMI response) | All | CMI |
| 2100.a | Humoral immune response results not available | All | HUM |
| 2100.b | CMI response results not available | All | CMI |
| 2120.a | Obvious incoherence or abnormality or error in data (data on humoral immune response) | All | HUM |
| 2120.b | Obvious incoherence or abnormality or error in data (data on CMI response) | All | CMI |

Note: CMI elimination codes are applicable only to subjects belonging to the CMI sub-cohort.

## 4.2.5. Elimination from unsolicited and solicited safety set

## 4.2.5.1. Excluded subjects

#### 4.2.5.1.1. Unsolicited safety set

Code 1030.b (not administering any NTHi-Mcat vaccine), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1150 (no post-vaccination safety data) will be used to identify subjects eliminated from the unsolicited safety set.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

Code 1150 will be attributed to subjects if <u>all</u> the following conditions are met: subject did not complete the safety assessment following the 7-day follow-up period after NTHi-Mcat vaccinations (i.e. phone contacts), did not return the pDiary, did not return for the scheduled visit 30-days after the NTHi-Mcat vaccinations and did not report any unsolicited AE.

## 4.2.5.1.2. Solicited safety set

Code 1030.b (not administering any NTHi-Mcat vaccine), code 800 (fraudulent data) and code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data) will be used to identify subjects eliminated from the solicited safety set.

## 5. STATISTICAL ANALYSES

Note that standard data derivation rules and statistical methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and statistical methods will be described in Section 9.

## 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (including age at first study vaccination in years, gender, race, ethnicity and smoking status) will be summarized by study groups and overall, using descriptive statistics:

- Frequency tables will be generated for categorical variables such as smoking status.
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age, height and weight.

Withdrawal status will be summarized by group using descriptive statistics:

- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal
- The number of subjects enrolled into the study as well as the number of subjects excluded from the PPS and mFAS will be tabulated.

#### 5.1.2. Additional considerations

Summaries of demographic/baseline characteristics will include: age, country, centre, gender, race, ethnicity, smoking status, pack-years and vital signs (including body mass index [BMI]).

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# 5.2. Exposure

# 5.2.1. Analysis of exposure planned in the protocol

None.

#### 5.2.2. Additional considerations

The number and percentage of subjects who received study vaccine doses will be tabulated for each study group (based on the ES).

# 5.3. Immunogenicity

# 5.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the PPS. A supplementary analysis may be based on the mFAS.

| Endpoint | Statistical analysis methods |
|---|---|
| Primary | Between group assessment Considering the sampling timepoint at 1 month after Dose 2 of NTHi-Mcat vaccine, the 2-sided 95% CIs for the group GMC ratio (Sh_NTHi-Mcat_1; _3; _6 group over NTHi-Mcat group) of anti-PD, anti-PE, anti-PilA, anti-UspA2 will be computed using an analysis of covariance (ANCOVA) model on the logarithm10 transformation of the concentrations. The ANCOVA model will include study group, smoking status (current or former), age category (50–59, 60–69, 70–80 years of age) and centre as factors and the antibody concentration before Dose 1 as covariate. |
| | Non-inferiority for a specific time-lag will be claimed if the lower limit of the 2-sided 95% CI for the GMC ratio will be above 0.667 for all anti-PD, anti-PE, anti-PiIA, anti-UspA2. The sequential procedure for multiple time-lags will be used: starting from the 6-months lag, the 3-months NI will be tested only if the 6-months NI will be demonstrated, while the 1-month NI will be tested only if the 6-months and 3-months NI will be both demonstrated. |
| Secondary - humoral | Within group assessment For each study group, for each sampling timepoint and for each antigen, the following statistics will be computed: Seropositivity rates with exact 95% CI (seropositivity defined using the assay lower limits of quantification [LLOQ]) Adjusted and unadjusted GMCs with 95% CI (adjustment by ANCOVA model, as specified above) The range and distribution of antibody concentrations The distribution of antibody concentrations for each antigen will be displayed using reverse cumulative distribution curves. |
| Secondary –cell-<br>mediated immune<br>response | CMI response induced by the NTHi-Mcat candidate vaccine will be evaluated, presenting the frequencies of antigen-specific CD4+ T cells per 10 <sup>6</sup> cells. The specific CD4+ T cells being identified as the CD4 + T cells expressing at least 2 different markers among CD40 Ligand (CD40L), IL-2, TNF- α, IFN- γ, IL-13 and IL-17 upon in vitro stimulation. Descriptive statistics (Min, Q1, Median, Mean, Q3 & Max) will be reported for each group at pre-Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh-NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of |

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

| Endpoint | Statistical analysis methods |
|---|---|
| | NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group). |
| Tertiary –cell-<br>mediated immune<br>response | <ul> <li>CMI response induced by the NTHi-Mcat candidate vaccine will be evaluated, presenting the frequencies of antigen-specific CD8+T cells per 10<sup>6</sup> cells. The specific CD8+T cells being identified as the CD8+ T cells expressing at least 2 different markers among CD40L, IL-2, TNF- α, IFN- γ, IL-13 and IL-17 upon in vitro stimulation.</li> <li>CMI response as the frequencies of specific CD4+/CD8+ T cells per 10<sup>6</sup> cells expressing any combination of cytokines/activation markers will be determined. The T-helper profile of the specific T-cell response in T-helper 1, T-helper 2 and T-helper 17 based on the specific expression of respectively IFN-γ, IL-13 and IL-17 will be characterized.</li> <li>Descriptive statistics (Min, Q1, Median, Mean, Q3 &amp; Max) will be reported for each group at pre-Dose 1 of the NTHi-Mcat investigational vaccine (Day 91; Day 151; Day 241 in the Sh-NTHi-Mcat groups and Day 1 in the NTHi-Mcat group), and 1 month after Dose 2 of NTHi-Mcat investigational vaccine (Day 181; Day 241; Day 331 in the Sh_NTHi-Mcat groups and Day 91 in the NTHi-Mcat group).</li> </ul> |

### 5.3.2. Additional considerations

The supplementary analysis based on the mFAS will be performed if the percentage of mFAS subjects excluded from the PPS is more than 10%.

#### 5.3.2.1. Analysis of humoral response

## Hypothesis related to the primary objective

The global null hypothesis related to the primary objective of the study is that at least 1 GMC ratio (Sh\_NTHi-Mcat over NTHi-Mcat) among anti-PD, anti-PE, anti-PilA, anti-UspA2 is inferior or equal to 0.667 in all time-lags under investigation at 1 month post-Dose 2 of NTHi-Mcat vaccine. This must be rejected in favour of the alternative hypothesis that all 4 GMCs (anti-PD, anti-PE, anti-PilA, anti-UspA2) are non-inferior in at least one time-lag group. Family-wise type I error is fixed at 2.5% (1-sided).

#### Geometric mean concentration and geometric mean concentration ratio

For each antigen and study group, at 1 month after Dose 2 of NTHi-Mcat vaccine, adjusted GMCs and GMCs ratios with corresponding 95% CIs will be obtained exponentiating (base 10) the least square means and the lower and upper limits of the 95% CIs derived from the ANCOVA model. The ANCOVA model will be implemented in SAS, similarly to the following code:

```
PROC GLM data=<dataset>;
BY antigen;
class group age smoking_status centre;
MODEL log(concentr) = group age smoking_status centre log(pre_concentr);
LSMEAN group / CL PDIFF ALPHA=0.05;
RUN;
```

Contrasts to be included: Sh\_NTHi-Mcat\_6 vs NTHi-Mcat, Sh\_NTHi-Mcat\_3 vs NTHi-Mcat, Sh\_NTHi-Mcat\_1 vs NTHi-Mcat.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

In addition, unadjusted GMCs and GMRs will be presented for each timepoint (pre-Dose 1 and post-Dose 2 of NTHi-Mcat vaccine) with a descriptive purpose.

## Permutation test (sensitivity analysis on primary objectives)

Based on the covariate-adaptive treatment assignment algorithm (see Section 10.3), the following permutation test will be performed as a sensitivity analysis on the primary objectives [Wiens, 2006, Hasegawa, 2009 and Ernst, 2004] in the PPS.

For each antigen, let  $\mathbf{X}$ =( $X_1$ , ...,  $X_N$ ) the logarithmically-transformed antibody concentrations for the NTHi-Mcat group and  $\mathbf{Y}_{1/3/6}$ =( $Y_1$ , ...,  $Y_N$ ) the logarithmically-transformed antibody concentrations for one of the Sh\_NTHi-Mcat groups at 1 month after Dose 2 of NTHi-Mcat vaccine, a non-inferiority permutation test can be obtained from a superiority permutation test on  $\dot{\mathbf{X}}$ =( $X_1$ , ...,  $X_N$ ) against  $\dot{\mathbf{Y}}_{1/3/6}$ =( $Y_1$  +  $\delta$ , ...,  $Y_N$  +  $\delta$ ) with  $\delta$  = 0.176 = -log<sub>10</sub>(0.667).

The original treatment assignment algorithm will be used to re-randomize subjects belonging to the NTHi-Mcat group and, individually, each of the Sh\_NTHi-Mcat groups (see step 2a) while keeping antibody concentrations, covariates and entry order as observed. This is in line with the experimental design comparing individually 3 treatment groups with a unique control group. The procedure will be as follows:

- 1. Fit the ANCOVA model to obtain the test statistics  $T^*_{1/3/6}$  for the superiority of  $\dot{\mathbf{X}}$  against  $\dot{\mathbf{Y}}_{1/3/6}$ .
- 2. For each of the Sh\_NTHi-Mcat\_k groups [k=1, 3, 6], estimate the distribution of the corresponding test statistics with R=10000 repetitions of the following 2 steps:
  - a. Re-randomize treatment assignment of groups  $\dot{\mathbf{X}}$  and  $\dot{\mathbf{Y}}_k$  alone (original algorithm), while keeping the remaining 2 groups fixed.
  - b. Re-fit the full ANCOVA model to re-obtain the test statistics  $T_k$
- 3. Derive the permutation p-values associated to the observed test statistics (from step 1) based on the empirical distributions in Step 2

$$\mathbf{p}_{1/3/6} = \mathbf{M} + 1/\mathbf{R} + 1$$

Where M is the number of repetitions such that  $T_{1/3/6} \ge T^*_{1/3/6}$ .

### Seropositivity rate and fold increase

For each antigen, timepoint and study group, the seropositivity rate (defined as the proportion of subjects with an antibody concentration greater or equal to the assay cutoff) with exact 95% CIs will be computed using the method referenced in section 10.1.5.1. Assay cut-offs are reported in section 9.1.1. In addition, percentages of subjects with a 2/4/8-fold increase will be presented with associated 95% CI.

#### **Reverse cumulative distribution curves**

Reverse cumulative distribution (RCD) curves for antibody concentrations will be plotted: the x-axis represents the antibody concentrations value (log-10 scale), while the

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

y-axis the percentage of subjects having a log-transformed antibody value greater or equal to the corresponding x-value.

## 5.3.2.2. Analysis of CMI response

The frequency of **antigen-specific** CD4+ or CD8+ T-cells for each individual subject is calculated as the difference between the frequency of CD4+ or CD8+ T-cells producing at least 2 activation markers among CD40 Ligand (CD40L), IL-2, TNF-  $\alpha$ , IFN-  $\gamma$ , IL-13 and IL-17, upon *in vitro* stimulation with the antigen (induction condition) minus the frequency of CD4+ or CD8+ T-cells producing at least 2 activation markers upon in vitro stimulation in medium only (background condition). For descriptive statistics purposes, differences less or equal to zero (0) are imputed to 1.

# 5.4. Analysis of safety and reactogenicity

## 5.4.1. Analysis of safety and reactogenicity planned in the protocol

All safety analyses will be performed on the solicited safety set, unsolicited safety set and exposed set.

| Endpoint | Statistical analysis methods |
|---|---|
| Secondary | Within group assessment The percentage of subjects with at least 1 local adverse event (AE) (solicited and unsolicited), with at least 1 general AE (solicited and unsolicited) and with any AE during the 7-days solicited follow-up period and the 30-days follow-up period will be tabulated by group with exact 95% CI after each NTHi-Mcat vaccine dose and overall. The percentage of NTHi-Mcat doses followed by at least 1 local AE (solicited and unsolicited), by at least 1 general AE (solicited and unsolicited) and by any AE will be tabulated by group with exact 95% CI. The same calculations will be performed for AEs rated as Grade 3, for AEs causally related to vaccination and Grade 3 AEs causally related to vaccination. |
| | The percentage of subjects reporting each individual solicited local and general AE during the 7-days solicited follow-up period after each dose of NTHi-Mcat vaccine will be tabulated by group with exact 95% CI. The percentage of NTHi-Mcat doses followed by each individual solicited local and general AE will be tabulated by group with exact 95% CI. Fever will be reported per 0.5°C cumulative increments. For all solicited symptoms, the same tabulation will be performed for Grade 3 AEs. |
| | The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) Dictionary for Adverse Event Terminology. The percentage of subjects with at least 1 report of unsolicited adverse event classified by the MedDRA and reported up to 30 days after NTHi-Mcat vaccinations will be tabulated by group with exact 95% CI. The same tabulation will be performed for Grade 3 unsolicited adverse events, for unsolicited adverse events with a causal relationship to vaccination and for Grade 3 AEs causally related to vaccination. |
| | The number of subjects who experienced any serious adverse event (SAE) or any potential immune-mediated disease (pIMD) from Day 1 to Day 331 and from Day 331 to Day 661 will be reported. |
| | The number of subjects who experienced any AE leading to study withdrawal, from first vaccination up to study conclusion, or any SAE related to study participation or concurrent GSK medication/vaccination, during the entire study period, will be reported. |
| | A summary of subjects reporting concomitant medication/product will be provided. |

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

#### 5.4.2. Additional considerations

## 5.4.2.1. Analysis of solicited AEs

The analysis of solicited AEs will be performed on the Solicited safety set.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals as follows:

- 0: <20 mm diameter
- 1:  $\geq$ 20 mm to  $\leq$ 50 mm diameter
- 2: >50 mm to  $\leq$ 100 mm diameter
- 3. > 100 mm diameter

Temperature (i.e. fever) will be scored at GSK Biologicals as follows:

- 0: <37.5°C
- 1: 37.5°C to 37.9°C
- 2: 38.0°C to 38.9°C
- 3: ≥39.0°C

Fever, defined as a body temperature of  $\geq$ 37.5°C irrespective of route of measurement, will be integrated to the summaries as a general AE.

In addition, body temperature will be broken down by 0.5°C increments:

- <36.0
- -36.0-36.4
- -36.5 36.9
- -37.0-37.4
- -37.5-37.9
- -38.0 38.4
- -38.5 38.9
- -39.0-39.4
- -39.5 39.9
- >40.0

Compliance of subjects in completing solicited AEs information will be reported as the percentage of subjects completing at least 80% of the diary entries related to local and general solicited AEs.

## 5.4.2.2. Analysis of unsolicited AEs

The analysis of unsolicited AEs will be performed on the Unsolicited safety set.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

Analysis of unsolicited AEs will be also stratified on AEs with a causal relationship to NTHi-Mcat vaccination.

## 5.4.2.3. Combined analysis of solicited and unsolicited AEs

The combined analysis of solicited and unsolicited AEs will be performed on the Unsolicited safety set.

Solicited AEs will be coded by MedDRA as per the following codes:

| Solicited symptom | Preferred Term code | Corresponding Preferred Term |
|---|---|---|
| | | decode |
| Pain | 10022086 | Injection site pain |
| Redness | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Gastrointestinal symptoms | 10017944 | Gastrointestinal disorder |
| Myalgia | 10028411 | Myalgia |
| Chills | 10008531 | Chills |
| Fever | 10037660 | Pyrexia |

Combined analysis of solicited and unsolicited AEs will be also stratified on AEs with a causal relationship to NTHi-Mcat vaccination (all solicited AEs are considered causally related).

## 5.4.2.4. Analysis of SAEs and pIMDs

The analysis of SAEs and pIMDs will be performed on the Exposed Set (ES).

Analysis of SAEs will include:

- All SAEs from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661
- Fatal SAEs from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
- Related SAEs:
  - To any study vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.
  - To the NTHi-Mcat vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661, from the day of the first NTHi-Mcat vaccination up to 1 month following the second dose, from the day of the first NTHi-Mcat vaccination up to 6 months following the second dose and from the day of the first NTHi-Mcat vaccination up to 12 months following the second dose (all groups except "Shingrix only").
  - To *Shingrix* vaccine, from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661 (all groups except NTHi-Mcat).

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

Analysis of pIMDs will include all occurrences from Day 1 to Day 331, from Day 331 to Day 661 and from Day 1 to Day 661.

## 5.4.2.5. Other safety analyses

Medications will be coded using GSKDRUG dictionary.

All collected concomitant medications and vaccinations will be listed. In case of pregnancies during the study, follow-up data and pregnancy outcomes will be described in detail.

#### 6. ANALYSIS INTERPRETATION

Except for analysis on primary objectives, with predefined success criteria and an appropriate type I error control, comparative analyses are descriptive with the aim to characterize the difference between groups.

With respect to confirmatory analyses on primary objectives the interpretation will be done in a hierarchical manner.

Each objective can only be reached if all the associated criteria are met and all previous objectives have been reached (see Figure 2): starting from the 6-months lag, the 3-months NI can be achieved only if the 6-months NI is demonstrated, while the 1-month NI can be achieved only if the 6-months and 3-months NI are both demonstrated.

This sequential procedure enables to control the overall type I error below 2.5% (one-sided) [Dmitrienko, 2009].

Figure 2 Sequence for evaluating the primary objective in order to control the overall type I error below 2.5% (one-sided)



209538 (NTHI MCAT-009) Statistical Analysis Plan Final

## 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

The integrated clinical study report (CSR) will contain at least the final analyses of all primary and secondary endpoints. If the data for tertiary endpoints become available at a later stage, (an) additional analysis/analyses will be performed. These analyses will be documented in annex(es) to the study report.

The analyses will be performed stepwise:

- A final analysis of immunogenicity, safety and reactogenicity for all subjects up to and including Day 331 ('Epoch 001') will be performed in a first step.
  - A complete study report containing all data of 'Epoch 001' will be written and made available to the investigators at this stage.
- Analysis conducted on the data collected for all subjects from Day 331 up to and including Day 661 ('Epoch 002') will be performed in a second step.

An integrated CSR containing all data from Epoch 001 and Epoch 002 will be written and made available to the investigators.

| Description | Disclosure Purpose<br>(CTRS=public posting, SR=study report, internal) |
|---|---|
| Final Analysis Epoch 001 | Web disclosure (CTRS), Study report (SR) |
| Analysis of Follow-up Epoch | Web disclosure (CTRS), Study report (SR) |

# 7.2. Statistical considerations for interim analyses

No interim analysis is planned for this study. Data up to and including Day 331 are considered 'final' and completed data, while the remaining safety data are considered long-term safety follow-up.

#### 8. CHANGES FROM PLANNED ANALYSES

Not applicable

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in Section 10.1

### 9.1. Data derivation

## 9.1.1. Assay cut-offs for serology results

| Component | Method | Unit <sup>1</sup> | Assay cut-off <sup>1</sup> |
|---|---|---|---|
| anti-PD antibody | ELISA | EU/mL | 153 |
| anti-PE antibody | ELISA | EU/mL | 25 |
| anti-PilA antibody | ELISA | EU/mL | 16 |
| anti-UspA2 IgG antibody | ELISA | EU/mL | 38 |

ELISA = Enzyme Linked Immunosorbent Assay; EU/ml = ELISA unit per millilitre; Ig = immunoglobulin; PD = protein D; from NTHi; PE = protein E from NTHi; PilA = type IV pili subunit from NTHi; UspA2 = ubiquitous surface protein A2 from Mcat

# 9.1.2. Attributing subjects to time-lag groups

For the purpose of safety analyses, the following rule will be used to attribute exposed subjects to a specific group.

- If a subject receives no *Shingrix* vaccination → NTHi-Mcat group
- If a subject receives at least 1 Shingrix vaccination, but no NTHi-Mcat vaccination
   → "Shingrix only" group
- If a subject receives at least 1 *Shingrix* vaccination and at least 1 NTHi-Mcat vaccination, the difference, in days, between the latest Shingrix vaccination and the earliest NTHi-Mcat vaccination will be computed and converted in months (diff):
  - diff  $\leq 2 \rightarrow$  Sh NTHi-Mcat 1 group
  - $2 < diff \le 4.5 \rightarrow Sh_NTHi-Mcat_3 group$
  - diff  $> 4.5 \rightarrow$  Sh NTHi-Mcat 6 group

#### 9.2. Statistical Method

Not applicable

<sup>1</sup> Assay cut-off and unit might be subject to change during the course of the study (e.g. in case of assay reoptimization, qualification, (re)validation or standardization). In this case, this will be documented in the clinical study report.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

#### 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in Section 9 (additional study-specific rules).

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the eCRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30th.

The following exceptions apply:

- Adverse event start dates with missing day:
  - If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that month.

#### 209538 | Statistical Analysis Plan | 01 Apr 2019 | TMF-855396 | 2.0

#### CONFIDENTIAL

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

- Adverse event start dates with missing day and month:
  - If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

## 10.1.2.3. Daily recording of solicited symptoms

#### 10.1.2.3.1. Studies with paper diaries

Denominators for the summary of local (or general) solicited symptoms will be calculated using the number of subjects who respond "Yes" or "No" to the question concerning the occurrence of local (or general) symptoms.

When a specific symptom is marked as having not occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=N for the specified post-vaccination period for the symptom in question), all daily measurements will be imputed as Grade 0.

When a specific symptom is marked as having occurred following a specific vaccination (i.e. SDTM CE.CEOCCUR=Y for the specified post-vaccination period for the symptom in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables

When the occurrence of a specific symptom is not present (i.e. SDTM CE.CEOCCUR is neither Y nor N for the specified post-vaccination period for the symptom in question) but the group of symptoms (local or general) is marked as having occurred (i.e. SDTM CE.CEOCCUR=Y), all missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the symptom summary tables.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

The following table shows how subjects contribute to each category for a specific solicited symptom over the Day X to Day Y post-vaccination period:

| Solicited symptom category | Subjects included in the calculation of the numerator |
|---|---|
| Any | All subjects with at least one occurrence of the symptom at Grade 1, Grade 2, or Grade 3 between Day X and Day Y or with the symptom marked as present and at least one missing daily recording between Day X and Day Y |
| At least grade 1 | All subjects with at least one occurrence of the symptom at Grade 1, Grade 2, or Grade 3 between Day X and Day Y |
| At least grade 2 | All subjects with at least one occurrence of the symptom at Grade 2 or Grade 3 between Day X and Day Y |
| At least grade 3 | All subjects with at least one occurrence of the symptom at Grade 3 between Day X and Day Y |

#### 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### 10.1.3. Data derivation

#### 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years

DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

## 10.1.3.2. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (weight in kilograms) / (height in meters) $^2$ 

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

## 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

## 10.1.3.4. Geometric mean concentrations (GMCs)

GMC calculations are performed by taking the inverse logarithm of the mean of the log-10 concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

#### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus 1 day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the symptom reported at Grade 1 or higher.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

## 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event eCRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.3.8. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarised, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study vaccines, an injection site reaction recorded for a subject following multiple vaccines will be counted as only one occurrence.

## 10.1.4. Display of decimals

## 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group
  - Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

## 10.1.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with 1 more decimal than the maximum number used to display the individual percentages, for example the difference between two percentages displayed with 1 decimal will be displayed with 2 decimals.

#### 10.1.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, BMI, pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height variables will be displayed with no decimals.

The maxima and minima of transformed weight variables will be displayed with no decimals with the exception of values below 10kg where 1 decimal will be displayed.

The maximum and minima of transformed body temperatures will be displayed with 1 decimal.

#### 10.1.4.4. Serological summary statistics

The number of decimals used when displaying GMCs and their confidence limits is shown in the following table:

| GMC value | Number of decimals to display |
|----------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the 1 with the higher number of decimals). For example, if GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

## 10.1.5. Statistical methodology

#### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

# 10.1.5.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Mietinnen and Nurminen [Miettinen, 1985].

#### 10.1.5.3. Adjusted GMC ratios

When between-group GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure.

#### 10.2. TFL ToC

The TFL ToC can be found in eTMF folder section 11.1.1.

# 10.3. Randomization method and minimization algorithm

The minimization algorithm used at the GSK internet randomization system (i.e. SBIR) for study NTHI MCAT-009 is based on the following reference: "White SJ, Freedman LS. Allocation of patients to treatment groups in a controlled clinical study. Br J Cancer 1978; 37: 849-857" [White, 1978] and it is described below:

#### **Notations**

- K=3 input values [Centre, Smoking status and Age category] to be used for minimization, each with a weight  $w_k=1$  (k=1,...,K) &  $l_k$  variants.
- I=4 treatment groups [NTHi-Mcat, Sh\_NTHi-Mcat\_6, Sh\_NTHi-Mcat\_3, Sh\_NTHi-Mcat\_1] with randomization ratio a<sub>1</sub>,...,a<sub>I</sub> [1:1:1:1]

#### Algorithm

For a new subject with input value variants  $s_1 ... s_K$ 

#### Step 1: Minimization computation

Step 1.1: Initialize Problem flag to 0

#### 209538 | Statistical Analysis Plan | 01 Apr 2019 | TMF-855396 | 2.0

#### CONFIDENTIAL

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

For each input value variant  $s_k$ , compute the number of subjects already enrolled in each treatment group.

Let  $b_{ik}$  the number for treatment i & input value variant  $s_k$ :  $b_{ik}$  is the total number of subjects already randomized (excluding subjects cancelled/withdrawn prior dose 1) in treatment i and with variant  $s_k$ .

Step 1.2: For each treatment i: compute  $A_i = 1/a_i * sum_k(w_k * b_{ik})$ 

Step 2: determine whether the algorithm is random or deterministic:

Generate R, a random number within [0-1], uniform distribution

Step 3: check determinism

If R < 0.9, go to step 4 (determinism) else go to step 5 (random)

Step 4: determinism

4.1: Identify all treatments with the lowest value A<sub>i</sub>

4.2: Select randomly one of the treatments identified in step 4.1, let it be T.

Go to step 6, if no more treatment then randomization failed

Step 5: randomization

Select randomly one of the treatments, let it be T.

Go to step 6, if no more treatment then randomization failed.

Step 6: treatment allocation

Assign one of the treatment nr. related to treatment T in the subject's center.

If no treatment nr. related to treatment T is available in the subject's center, then go & repeat step 4 (determinism) or 5 (random) while dropping treatment T (set problem flag=1).

209538 (NTHI MCAT-009) Statistical Analysis Plan Final

## 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

Dmitrienko, A., Tamhane, A. C., & Bretz, F. (2009). Multiple testing problems in pharmaceutical statistics. CRC press.

Ernst MD, Permutation Methods: A Basis for Exact Inference. *Statistical Science*, 2004; 19: 676-685.

Hasegawa T, Tango T. Permutation test Following Covariate-Adaptive Randomization in Randomized Controlled Trials. *Journal of Biopharmaceutical Statistics*, 2009; 19: 106-119.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. *Statistics in Medicine*, 1985;4:213-226.

White SJ, Freedman LS. Allocation of patients to treatment groups in a controlled clinical study. *Br J Cancer*, 1978;37: 849-857

Wiens BL, Randomization as basis for inference in noninferiority trials. *Pharmaceutical Statistics*, 2006; 5: 265-271